CLINICAL TRIAL: NCT00413660
Title: A Phase 2B, Randomized, Double Blind, Placebo-Controlled, Multicenter Study To Compare 6 Dose Regimens Of CP-690,550 Vs. Placebo, Each Combined With Methotrexate, Administered For 6 Months In The Treatment Of Subjects With Active Rheumatoid Arthritis Who Have Had An Inadequate Response To Methotrexate Alone
Brief Title: Comparison Of 6 CP-690,550 Doses Vs.Placebo, Each Combined With Methotrexate, For The Treatment Of Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921025
Record Dates: First submitted 2006-12-18; First posted 2006-12-20 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: DMARD therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- CP 690,550 1 mg BID (Experimental)
  Interventions: Drug: CP-690,550
- CP 690,550 10 mg BID (Experimental)
  Interventions: Drug: CP-690,550
- CP 690,550 15 mg (Experimental)
  Interventions: Drug: CP-690,550
- CP 690,550 3 mg BID (Experimental)
  Interventions: Drug: CP-690,550
- CP 690,550 5 mg BID (Experimental)
  Interventions: Drug: CP-690,550
- CP-690,550 20 mg QD (Experimental)
  Interventions: Drug: CP-690,550
- Placebo (Placebo Comparator): Dummy tablets
  Interventions: Other: placebo

INTERVENTIONS:
Drug: CP-690,550 — 4 blinded tablets administered BID
  Arms: CP 690,550 1 mg BID
Drug: CP-690,550 — 4 blinded tablets administered BID
  Arms: CP 690,550 10 mg BID
Drug: CP-690,550 — 4 blinded tablets administered BID
  Arms: CP 690,550 15 mg
Drug: CP-690,550 — 4 blinded tablets administered BID
  Arms: CP 690,550 3 mg BID
Drug: CP-690,550 — 4 blinded tablets administered BID
  Arms: CP 690,550 5 mg BID
Drug: CP-690,550 — Oral tablets
  Arms: CP-690,550 20 mg QD
Other: placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness and safety, over 6 months, of 6 dose regimens of CP-690,550, combined with methotrexate, for the treatment of adults with active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis
* Inadequate response to stably dosed methotrexate

Exclusion Criteria:

* Current therapy with any DMARD or biologic other than methotrexate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (68):
- United States (29):
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, DeBary, Florida
  - Pfizer Investigational Site, Lake Mary, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Zephyrhills, Florida
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Binghamton, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Philladelphia, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Mesquite, Texas
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Onalaska, Wisconsin
- Argentina (2):
  - Pfizer Investigational Site, Capital Federal, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
- Brazil (3):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Sofia, Bulgaria
- Chile (4):
  - Pfizer Investigational Site, Viña del Mar, Región de Valparaíso
  - Pfizer Investigational Site, Providencia, RM
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Santiago, Santiago Metropolitan
- Czechia (5):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Praha 11 - Chodov
  - Pfizer Investigational Site, Zlín
- Hungary (4):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Komárom
  - Pfizer Investigational Site, Szolnok
  - Pfizer Investigational Site, Veszprém
- Mexico (2):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Morelia, Michoacán
- Poland (6):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Grudziądz
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Sopot
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Slovakia (3):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Piešťany
  - Pfizer Investigational Site, Žilina
- Spain (4):
  - Pfizer Investigational Site, Santiago de Compostela, A Coruña
  - Pfizer Investigational Site, Guadalajara, Guadalajara
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla
- Sweden (2):
  - Pfizer Investigational Site, Jönköping
  - Pfizer Investigational Site, Umeå
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Mariette X, Chen C, Biswas P, Kwok K, Boy MG. Lymphoma in the Tofacitinib Rheumatoid Arthritis Clinical Development Program. Arthritis Care Res (Hoboken). 2018 May;70(5):685-694. doi: 10.1002/acr.23421. Epub 2018 Apr 2. PMID 28941219
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Wallenstein GV, Kanik KS, Wilkinson B, Cohen S, Cutolo M, Fleischmann RM, Genovese MC, Gomez Reino J, Gruben D, Kremer J, Krishnaswami S, Lee EB, Pascual-Ramos V, Strand V, Zwillich SH. Effects of the oral Janus kinase inhibitor tofacitinib on patient-reported outcomes in patients with active rheumatoid arthritis: results of two Phase 2 randomised controlled trials. Clin Exp Rheumatol. 2016 May-Jun;34(3):430-42. Epub 2016 Apr 28. PMID 27156561
- [Derived] Charles-Schoeman C, Burmester G, Nash P, Zerbini CA, Soma K, Kwok K, Hendrikx T, Bananis E, Fleischmann R. Efficacy and safety of tofacitinib following inadequate response to conventional synthetic or biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2016 Jul;75(7):1293-301. doi: 10.1136/annrheumdis-2014-207178. Epub 2015 Aug 14. PMID 26275429
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- [Derived] Kremer JM, Cohen S, Wilkinson BE, Connell CA, French JL, Gomez-Reino J, Gruben D, Kanik KS, Krishnaswami S, Pascual-Ramos V, Wallenstein G, Zwillich SH. A phase IIb dose-ranging study of the oral JAK inhibitor tofacitinib (CP-690,550) versus placebo in combination with background methotrexate in patients with active rheumatoid arthritis and an inadequate response to methotrexate alone. Arthritis Rheum. 2012 Apr;64(4):970-81. doi: 10.1002/art.33419. Epub 2011 Oct 17. PMID 22006202
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921025&StudyName=Comparison%20Of%206%20CP-690%2C550%20Doses%20Vs.Placebo%2C%20Each%20Combined%20With%20Methotrexate%2C%20For%20The%20Treatment%20Of%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 1 mg: CP-690,550 1 milligram (mg) tablet orally twice daily for 24 weeks. Participants who failed to achieve a minimum improvement of at least 20 percent (%) reduction in both swollen and tender joint counts over baseline at Week 12 visit were reassigned to CP-690,550 1 mg to 5 mg (R) treatment arm for next 12 weeks.
- CP-690,550 3 mg: CP-690,550 3 mg tablet orally twice daily for 24 weeks. Participants who failed to achieve a minimum improvement of at least 20% reduction in both swollen and tender joint counts over baseline at Week 12 visit were reassigned to CP-690,550 3 mg to 5 mg (R) treatment arm for next 12 weeks.
- CP-690,550 5 mg: CP-690,550 5 mg tablet orally twice daily for 24 weeks.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily for 24 weeks.
- CP-690,550 15 mg: CP-690,550 15 mg tablet orally twice daily for 24 weeks.
- CP-690,550 20 mg: CP-690,550 20 mg tablet orally once daily as morning dose and matching placebo tablet orally once daily as evening dose for 24 weeks. Participants who failed to achieve a minimum improvement of at least 20% reduction in both swollen and tender joint counts over baseline at Week 12 visit were reassigned to CP-690,550 20 mg to 5 mg (R) treatment arm for next 12 weeks.
- Placebo: Matching placebo tablet orally twice daily for 24 weeks. Participants who failed to achieve a minimum improvement of at least 20 % reduction in both swollen and tender joint counts over baseline at Week 12 visit were reassigned to Placebo to CP-690,550 5 mg (R) treatment arm for next 12 weeks.
- CP-690,550 1 mg to CP-690,550 5 mg (R): Participants who failed to achieve minimum improvement in CP-690,550 1 mg treatment arm, after Week 12 visit received CP-690,550 5 mg tablet orally twice daily up to Week 24.
- CP-690,550 3 mg to CP-690,550 5 mg (R): Participants who failed to achieve minimum improvement in CP-690,550 3 mg treatment arm, after Week 12 visit received CP-690,550 5 mg tablet orally twice daily up to Week 24.
- CP-690,550 20 mg to CP-690,550 5 mg (R): Participants who failed to achieve minimum improvement in CP-690,550 20 mg treatment arm, after Week 12 visit received CP-690,550 5 mg tablet orally twice daily up to Week 24.
- Placebo to CP-690,550 5 mg (R): Participants who failed to achieve minimum improvement in placebo treatment arm, after Week 12 visit received CP-690,550 5 mg tablet orally twice daily up to Week 24.
Period: Up To Week 12
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | Placebo | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo to CP-690,550 5 mg (R)
Started | 71 | 68 | 71 | 75 | 75 | 80 | 69 | 0 | 0 | 0 | 0
Treated | 70 | 68 | 71 | 74 | 75 | 80 | 69 | 0 | 0 | 0 | 0
Completed | 64 | 61 | 64 | 67 | 66 | 70 | 58 | 0 | 0 | 0 | 0
Not Completed | 7 | 7 | 7 | 8 | 9 | 10 | 11 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 1 | 4 | 6 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Randomized, Not Treated | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 3 | 1 | 6 | 1 | 2 | 4 | 3 | 0 | 0 | 0 | 0
Period: Post Week 12
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | Placebo | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo to CP-690,550 5 mg (R)
Started | 43 | 48 | 64 | 67 | 66 | 57 | 40 | 21 | 13 | 13 | 18
Completed | 40 | 44 | 56 | 66 | 60 | 54 | 37 | 21 | 13 | 12 | 17
Not Completed | 3 | 4 | 8 | 1 | 6 | 3 | 3 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 2 | 0 | 2 | 1 | 4 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 1 | 2 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CP-690,550 1 mg: CP-690,550 1 mg tablet orally twice daily for 24 weeks. Participants who failed to achieve a minimum improvement of at least 20% reduction in both swollen and tender joint counts over baseline at Week 12 visit were reassigned to CP-690,550 1 mg to 5 mg (R) treatment arm for next 12 weeks.
- Total: Total of all reporting groups
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | Placebo | Total
Number analyzed (Participants) | 70 | 68 | 71 | 74 | 75 | 80 | 69 | 507
Age, Customized [Number; unit: participants]
  18 to 44 Years | 15 | 23 | 19 | 9 | 14 | 15 | 17 | 112
  45 to 64 Years | 47 | 31 | 42 | 49 | 49 | 49 | 40 | 307
  Greater Than or Equal to (>=) 65 Years | 8 | 14 | 10 | 16 | 12 | 16 | 12 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 52 | 57 | 55 | 66 | 63 | 56 | 406
  Male | 13 | 16 | 14 | 19 | 9 | 17 | 13 | 101

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR20 response: >= 20% improvement in tender joints count (TJC); >= 20% improvement in swollen joints count (SJC); and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 12
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study treatment. Missing values were imputed using Baseline Observation Carried Forward (BOCF).
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 71 | 74 | 75 | 80 | 69
percentage of participants | 47.14 | 55.88 | 56.34 | 58.11 | 56.00 | 56.25 | 36.23

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: >= 20% improvement in TJC; >= 20% improvement in SJC; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, 4, 6, 8, 16, 20, 24/Early Termination (ET)
Population: FAS included all randomized participants who received at least 1 dose of study treatment. Missing values were imputed using BOCF. Here "n" is number of participants evaluable at specific time points for each arm group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 80 | 13 | 69 | 18
percentage of participants
  Week 2 (n=70,0,68,0,71,74,75,80,0,69,0) | 21.43 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.76 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.99 | 31.08 | 40.00 | 33.75 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.94 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=70,0,68,0,71,74,75,80,0,69,0) | 37.14 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.59 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.48 | 45.95 | 54.67 | 51.25 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 24.64 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=70,0,68,0,71,74,75,80,0,69,0) | 44.29 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 54.41 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 57.75 | 55.41 | 56.00 | 50.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.68 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=70,0,68,0,71,74,75,80,0,69,0) | 50.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 54.41 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 54.93 | 56.76 | 64.00 | 56.25 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.33 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=49,21,55,13,71,74,75,67,13,51,18) | 63.3 | 0.0 | 60.0 | 0.0 | 53.5 | 64.9 | 62.7 | 64.2 | 0.0 | 43.1 | 0.0
  Week 20 (n=49,21,55,13,71,74,75,67,13,51,18) | 59.2 | 0.0 | 67.3 | 0.0 | 57.7 | 62.2 | 61.3 | 64.2 | 0.0 | 47.1 | 0.0
  Week 24 (n=49,21,55,13,71,74,75,67,13,51,18) | 59.2 | 0.0 | 65.5 | 0.0 | 59.2 | 66.2 | 65.3 | 62.7 | 0.0 | 47.1 | 0.0

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: >= 50% improvement in TJC or SJC and 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 80 | 13 | 69 | 18
percentage of participants
  Week 2 (n=70,0,68,0,71,74,75,80,0,69,0) | 1.43 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.88 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.63 | 4.05 | 17.33 | 15.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.90 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=70,0,68,0,71,74,75,80,0,69,0) | 4.29 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.18 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.27 | 20.27 | 26.67 | 25.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.90 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=70,0,68,0,71,74,75,80,0,69,0) | 10.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 29.41 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.99 | 27.03 | 32.00 | 27.50 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.70 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=70,0,68,0,71,74,75,80,0,69,0) | 17.14 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.35 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.39 | 28.38 | 41.33 | 32.50 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.39 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=70,0,68,0,71,74,75,80,0,69,0) | 22.86 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 29.41 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.62 | 28.38 | 44.00 | 36.25 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.39 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=49,21,55,13,71,74,75,67,13,51,18) | 38.8 | 0.0 | 43.6 | 0.0 | 38.0 | 36.5 | 40.0 | 41.8 | 0.0 | 21.6 | 0.0
  Week 20 (n=49,21,55,13,71,74,75,67,13,51,18) | 38.8 | 0.0 | 45.5 | 0.0 | 38.0 | 40.5 | 48.0 | 47.8 | 0.0 | 31.4 | 0.0
  Week 24 (n=49,21,55,13,71,74,75,67,13,51,18) | 44.9 | 0.0 | 34.5 | 0.0 | 39.4 | 39.2 | 46.7 | 46.3 | 0.0 | 31.4 | 0.0

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: >= 70% improvement in TJC or SJC and 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 80 | 13 | 69 | 18
percentage of participants
  Week 2 (n=70,0,68,0,71,74,75,80,0,69,0) | 1.43 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.47 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.41 | 1.35 | 6.67 | 2.50 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=70,0,68,0,71,74,75,80,0,69,0) | 2.86 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.35 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.00 | 14.86 | 13.33 | 12.50 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.45 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=70,0,68,0,71,74,75,80,0,69,0) | 1.43 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.24 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.90 | 9.46 | 16.00 | 12.50 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.35 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=70,0,68,0,71,74,75,80,0,69,0) | 8.57 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 14.71 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.27 | 16.22 | 16.00 | 17.50 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.80 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=70,0,68,0,71,74,75,80,0,69,0) | 4.29 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 20.59 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 18.31 | 12.16 | 24.00 | 23.75 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.80 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=49,21,55,13,71,74,75,67,13,51,18) | 16.3 | 0.0 | 21.8 | 0.0 | 18.3 | 18.9 | 24.0 | 22.4 | 0.0 | 9.8 | 0.0
  Week 20 (n=49,21,55,13,71,74,75,67,13,51,18) | 20.4 | 0.0 | 29.1 | 0.0 | 23.9 | 24.3 | 28.0 | 28.4 | 0.0 | 13.7 | 0.0
  Week 24 (n=49,21,55,13,71,74,75,67,13,51,18) | 28.6 | 0.0 | 23.6 | 0.0 | 21.1 | 18.9 | 32.0 | 28.4 | 0.0 | 9.8 | 0.0

5. Secondary Outcome: Area Under the Numeric Index of American College of Rheumatology Response (ACR-n) Curve
Description: ACR-n: calculated for each participant by taking the lowest percentage improvement in (1) SJC or (2) TJC or (3) the median of the remaining 5 components of the ACR response (participant's assessment of disease activity; participant's global assessment of pain; physician's assessment of disease activity; participant's assessment of physical function; an acute phase reactant value - CRP). Negative numbers indicate worsening. The area under the curve (AUC) for ACR-n is the measure of the area under the curve of the mean change from baseline in ACR-n. The trapezoidal rule was used to compute the AUC.
Time Frame: Baseline up to Week 2, 4, 6, 8, 12
Population: FAS included all randomized participants who received at least 1 dose of study treatment. Missing values were imputed using Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | Placebo
Number analyzed (Participants) | 70 | 68 | 71 | 74 | 75 | 80 | 69
units on a scale
  Week 2 | -14.07 (247.36) | 22.16 (243.19) | 4.47 (319.92) | -21.34 (661.05) | 88.72 (287.91) | 36.55 (267.26) | -113.31 (429.17)
  Week 4 | 61.66 (622.43) | 163.40 (659.05) | 92.24 (919.49) | 7.29 (2038.26) | 341.52 (820.16) | 170.23 (825.49) | -296.38 (1270.69)
  Week 6 | 244.11 (948.25) | 442.29 (1087.57) | 348.96 (1446.07) | 111.83 (3626.48) | 716.69 (1285.36) | 402.21 (1428.69) | -453.18 (2265.12)
  Week 8 | 464.42 (1424.59) | 772.65 (1594.84) | 693.90 (1952.07) | 239.54 (5389.58) | 1154.14 (1733.13) | 725.67 (1954.96) | -571.99 (3310.17)
  Week 12 | 995.34 (2349.99) | 1511.40 (2711.76) | 1420.20 (3284.51) | 588.45 (8969.29) | 1974.18 (3231.70) | 1504.58 (2979.75) | -755.22 (5107.45)

6. Secondary Outcome: Tender Joints Count (TJC)
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: FAS included all randomized participants who received at least 1 dose of study treatment. Here "N" (number of participants analyzed) signifies participants evaluable for this measure and "n" signifies participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 80 | 12 | 69 | 17
tender joints
  Baseline (n=70,0,68,0,71,74,75,80,0,69,0) | 23.64 (11.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 22.79 (10.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 21.46 (12.95) | 24.84 (12.51) | 23.68 (12.71) | 23.11 (12.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 21.59 (13.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=68,0,68,0,68,73,73,79,0,66,0) | 18.62 (12.09) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.71 (11.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.56 (10.44) | 17.34 (12.13) | 16.32 (13.18) | 15.33 (12.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 18.86 (13.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,65,0,67,70,72,76,0,66,0) | 15.01 (11.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.80 (10.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.06 (11.59) | 14.01 (14.73) | 13.00 (12.48) | 13.75 (13.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.17 (12.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,65,0,69,71,72,74,0,62,0) | 14.48 (12.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.12 (9.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.23 (10.44) | 13.55 (14.38) | 11.51 (12.67) | 13.22 (13.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 14.74 (13.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,62,0,66,67,70,73,0,61,0) | 14.24 (12.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.18 (10.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.82 (11.08) | 12.22 (13.75) | 9.49 (11.71) | 11.15 (13.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.57 (14.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=64,0,59,0,64,66,66,70,0,61,0) | 12.84 (12.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.83 (9.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.09 (11.65) | 10.88 (12.79) | 10.18 (12.65) | 11.27 (13.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.77 (14.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,45,13,58,66,61,55,12,37,16) | 8.07 (9.11) | 19.33 (15.70) | 6.02 (7.97) | 19.15 (16.42) | 8.64 (12.25) | 9.77 (12.49) | 8.39 (11.32) | 7.07 (8.86) | 26.25 (19.07) | 8.51 (7.25) | 15.56 (18.52)
  Week 20 (n=39,21,44,13,57,66,59,55,12,37,17) | 8.08 (11.06) | 13.76 (12.02) | 5.32 (6.35) | 15.00 (11.47) | 7.16 (9.91) | 8.27 (11.32) | 6.98 (9.96) | 6.51 (10.55) | 23.00 (16.59) | 7.62 (7.26) | 15.24 (17.68)
  Week 24 (n=40,20,44,13,55,64,60,53,12,36,17) | 7.45 (10.88) | 14.80 (14.09) | 5.52 (5.65) | 13.92 (9.93) | 6.85 (9.51) | 8.20 (9.94) | 6.37 (8.72) | 5.87 (7.68) | 21.67 (13.69) | 5.33 (5.74) | 15.88 (17.46)

7. Secondary Outcome: Change From Baseline in Tender Joints Count (TJC) at Week 2, 4, 6, 8, 12, 16, 20 and 24/ET
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 68 | 21 | 68 | 13 | 68 | 73 | 73 | 79 | 12 | 66 | 17
tender joints
  Week 2 (n=68,0,68,0,68,73,73,79,0,66,0) | -4.68 (7.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.09 (9.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.06 (9.36) | -7.62 (8.48) | -7.68 (10.20) | -7.78 (9.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.27 (7.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,65,0,67,70,72,76,0,66,0) | -8.28 (8.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.26 (9.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.42 (9.73) | -10.77 (10.25) | -10.90 (11.13) | -9.59 (10.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.03 (10.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,65,0,69,71,72,74,0,62,0) | -8.86 (10.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.78 (10.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.01 (9.64) | -11.07 (9.94) | -12.14 (10.07) | -10.58 (9.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.69 (11.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,62,0,66,67,70,73,0,61,0) | -9.08 (10.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -12.69 (11.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.50 (9.06) | -11.93 (10.92) | -13.76 (11.73) | -12.26 (9.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.03 (13.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=64,0,59,0,64,66,66,70,0,61,0) | -10.67 (10.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -14.00 (12.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.88 (11.01) | -13.47 (9.96) | -14.24 (11.80) | -12.77 (10.92) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.84 (12.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,45,13,58,66,61,55,12,37,16) | -14.05 (9.97) | -6.81 (7.90) | -17.44 (10.54) | -1.00 (14.29) | -12.93 (12.63) | -14.58 (11.19) | -15.05 (11.31) | -15.65 (9.29) | -2.33 (15.69) | -10.16 (9.92) | -8.06 (10.88)
  Week 20 (n=39,21,44,13,57,66,59,55,12,37,17) | -13.64 (10.63) | -12.38 (10.61) | -18.36 (9.52) | -5.15 (11.07) | -14.58 (11.94) | -16.08 (10.43) | -16.64 (10.73) | -15.67 (9.33) | -5.58 (11.32) | -11.05 (11.86) | -8.24 (11.19)
  Week 24 (n=40,21,44,13,55,64,60,53,12,36,17) | -14.53 (10.83) | -10.40 (11.27) | -18.16 (9.82) | -6.23 (10.54) | -14.93 (11.72) | -16.36 (9.39) | -17.03 (10.39) | -16.36 (10.60) | -6.92 (12.62) | -13.17 (9.90) | -7.59 (12.39)

8. Secondary Outcome: Swollen Joints Count (SJC)
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 80 | 12 | 69 | 17
swollen joints
  Baseline (n=70,0,68,0,71,74,75,80,0,69,0) | 16.51 (8.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.68 (8.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 14.06 (7.44) | 14.74 (7.46) | 15.33 (7.02) | 15.21 (8.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.72 (8.83) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=68,0,68,0,68,73,73,79,0,66,0) | 12.62 (7.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.97 (9.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.51 (6.30) | 10.14 (7.92) | 10.07 (7.29) | 10.14 (6.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.41 (9.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,65,0,67,70,72,76,0,66,0) | 9.85 (7.74) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.58 (8.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.01 (7.45) | 7.53 (6.98) | 7.85 (6.70) | 8.61 (7.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.11 (8.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,65,0,69,71,72,74,0,62,0) | 8.77 (6.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.23 (7.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.22 (6.00) | 7.10 (7.62) | 6.60 (6.31) | 7.66 (7.43) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.39 (9.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,62,0,66,67,70,73,0,61,0) | 8.20 (7.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.63 (7.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.35 (5.03) | 6.78 (7.43) | 6.01 (6.22) | 7.22 (8.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.16 (8.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=64,0,59,0,64,66,66,70,0,61,0) | 8.31 (8.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.36 (6.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.13 (6.82) | 5.50 (5.84) | 4.85 (6.04) | 6.80 (8.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.79 (9.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,45,13,58,66,61,55,12,37,16) | 5.83 (7.43) | 8.90 (7.55) | 3.49 (3.78) | 10.00 (10.51) | 3.84 (4.40) | 4.74 (5.64) | 4.26 (5.40) | 3.58 (3.54) | 14.50 (12.99) | 5.97 (5.98) | 8.63 (7.70)
  Week 20 (n=39,21,44,13,57,66,59,55,12,37,17) | 4.95 (7.82) | 7.33 (8.75) | 3.36 (5.19) | 8.54 (9.85) | 3.95 (5.80) | 4.21 (5.59) | 3.27 (4.02) | 3.31 (4.19) | 12.25 (8.25) | 5.00 (6.65) | 7.41 (9.27)
  Week 24 (n=40,20,44,13,55,64,60,53,12,36,17) | 4.10 (4.83) | 8.65 (8.77) | 3.73 (5.35) | 7.00 (7.14) | 3.71 (4.33) | 4.41 (6.86) | 3.03 (3.75) | 2.89 (2.97) | 11.25 (9.81) | 4.11 (3.90) | 7.94 (8.90)

9. Secondary Outcome: Change From Baseline in Swollen Joints Count (SJC) at Week 2, 4, 6, 8, 12, 16, 20 and 24/ET
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 68 | 21 | 68 | 13 | 68 | 73 | 73 | 79 | 12 | 66 | 17
swollen joints
  Week 2 (n=68,0,68,0,68,73,73,79,0,66,0) | -3.43 (5.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.71 (7.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.24 (6.33) | -4.75 (5.57) | -5.45 (7.74) | -5.04 (7.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.12 (5.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,65,0,67,70,72,76,0,66,0) | -6.19 (6.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.25 (8.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.97 (5.44) | -7.34 (6.27) | -7.64 (6.77) | -6.74 (8.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.56 (5.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,65,0,69,71,72,74,0,62,0) | -7.41 (6.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.42 (9.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.68 (6.30) | -7.68 (7.35) | -8.68 (6.73) | -7.97 (7.54) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.48 (6.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,62,0,66,67,70,73,0,61,0) | -7.80 (8.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.03 (9.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.74 (6.94) | -8.06 (7.40) | -9.31 (7.51) | -8.26 (8.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.15 (6.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=64,0,59,0,64,66,66,70,0,61,0) | -7.61 (9.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.47 (9.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.13 (8.00) | -9.20 (7.16) | -10.68 (7.37) | -8.84 (8.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.52 (8.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,45,13,58,66,61,55,12,37,16) | -10.67 (8.78) | -5.95 (6.99) | -13.00 (8.90) | -2.46 (5.77) | -10.60 (7.43) | -9.95 (6.97) | -10.66 (6.75) | -10.65 (7.09) | -5.83 (13.62) | -8.65 (6.58) | -6.88 (6.51)
  Week 20 (n=39,21,44,13,57,66,59,55,12,37,17) | -10.95 (8.32) | -7.52 (8.20) | -13.36 (8.25) | -3.92 (5.72) | -10.39 (6.98) | -10.48 (7.21) | -11.61 (6.35) | -11.00 (6.99) | -8.08 (9.89) | -9.62 (7.31) | -7.88 (9.21)
  Week 24 (n=40,20,44,13,55,64,60,53,12,36,17) | -12.15 (7.83) | -6.60 (7.50) | -13.00 (8.52) | -5.46 (6.77) | -10.25 (6.70) | -10.48 (6.33) | -11.70 (6.38) | -11.57 (7.50) | -9.08 (11.99) | -10.28 (7.46) | -7.35 (6.47)

10. Secondary Outcome: Patient Assessment of Arthritis Pain
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) Visual Analog Scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 67 | 13 | 71 | 74 | 75 | 80 | 12 | 69 | 17
mm
  Baseline (n=70,0,66,0,71,74,75,80,0,69,0) | 59.96 (25.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 55.05 (24.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 54.87 (26.68) | 56.66 (25.42) | 55.83 (22.85) | 59.61 (23.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 51.19 (27.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=68,0,67,0,68,73,73,79,0,66,0) | 49.53 (24.99) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.33 (23.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.35 (24.31) | 41.26 (22.18) | 37.82 (22.17) | 40.57 (27.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.91 (25.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,65,0,67,70,72,76,0,66,0) | 45.57 (24.99) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.83 (22.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.03 (24.25) | 39.34 (25.09) | 35.81 (23.88) | 34.39 (24.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.02 (24.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,65,0,69,71,72,74,0,61,0) | 38.74 (24.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.75 (25.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.33 (24.18) | 34.38 (23.15) | 32.97 (23.50) | 33.65 (25.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.21 (27.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,62,0,66,67,70,73,0,61,0) | 38.97 (23.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 28.81 (23.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.55 (25.00) | 34.60 (24.04) | 30.26 (22.20) | 31.16 (24.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.34 (26.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=64,0,59,0,64,65,66,70,0,61,0) | 35.92 (22.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.90 (24.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 28.88 (22.80) | 33.78 (25.50) | 31.48 (24.86) | 31.09 (26.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.02 (26.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,45,13,58,66,61,54,12,37,16) | 27.83 (18.65) | 40.38 (21.81) | 29.67 (24.13) | 39.31 (24.13) | 28.98 (22.15) | 30.33 (22.04) | 27.07 (20.76) | 24.56 (23.46) | 51.25 (21.95) | 30.08 (22.81) | 38.38 (24.52)
  Week 20 (n=39,21,43,13,57,65,59,55,12,37,17) | 29.28 (22.75) | 35.71 (22.42) | 26.63 (23.48) | 42.31 (28.61) | 25.91 (23.10) | 33.66 (24.02) | 24.69 (20.98) | 24.58 (26.24) | 43.92 (27.07) | 25.08 (21.19) | 33.00 (27.70)
  Week 24 (n=40,20,44,13,55,63,60,53,12,36,17) | 25.53 (21.05) | 38.15 (26.27) | 25.98 (20.61) | 35.62 (28.27) | 24.45 (20.24) | 28.65 (21.11) | 24.47 (22.23) | 19.92 (18.27) | 35.33 (27.17) | 27.14 (21.17) | 33.65 (26.15)

11. Secondary Outcome: Change From Baseline in Patient Assessment of Arthritis Pain at Week 2, 4, 6, 8, 12, 16, 20 and 24/ET
Description: Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 68 | 21 | 65 | 13 | 68 | 73 | 73 | 79 | 12 | 66 | 17
mm
  Week 2 (n=65,0,68,0,68,73,73,79,0,66,0) | -9.49 (24.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.00 (20.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.76 (26.22) | -15.30 (25.46) | -17.67 (24.58) | -18.84 (25.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.55 (25.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,63,0,67,70,72,76,0,66,0) | -13.44 (26.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -17.11 (23.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -14.76 (24.06) | -17.80 (30.25) | -20.39 (28.95) | -24.74 (26.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.26 (28.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,63,0,69,71,72,74,0,61,0) | -19.56 (31.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -22.71 (28.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -21.07 (29.07) | -22.94 (29.71) | -22.61 (28.87) | -26.97 (26.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.61 (29.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,60,0,66,67,70,73,0,61,0) | -19.91 (26.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -26.23 (29.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -18.11 (29.71) | -21.84 (30.42) | -24.66 (30.16) | -29.08 (27.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.97 (28.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=64,0,57,0,64,65,66,70,0,61,0) | -23.16 (28.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -24.39 (30.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -25.75 (29.47) | -24.02 (27.96) | -23.95 (29.90) | -29.67 (28.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.30 (30.14) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,45,13,58,66,61,54,12,37,16) | -34.02 (31.75) | -13.48 (25.66) | -27.19 (24.93) | -15.15 (21.97) | -26.50 (28.81) | -26.64 (25.04) | -27.97 (29.32) | -32.09 (24.84) | -19.00 (29.73) | -17.22 (35.13) | -18.19 (21.36)
  Week 20 (n=39,21,41,13,57,65,59,55,12,37,17) | -31.54 (36.96) | -18.14 (25.06) | -32.37 (26.83) | -12.15 (25.36) | -29.54 (30.99) | -22.78 (30.27) | -30.97 (31.28) | -32.95 (27.48) | -26.33 (33.15) | -22.22 (30.68) | -21.82 (21.49)
  Week 24 (n=40,20,42,13,55,63,60,53,12,36,17) | -36.08 (32.62) | -15.40 (24.78) | -33.19 (25.68) | -18.85 (24.73) | -29.89 (30.87) | -28.51 (28.01) | -31.00 (31.88) | -36.98 (27.86) | -34.92 (31.74) | -21.08 (32.99) | -21.18 (26.30)

12. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS, where 0 mm = very well and 100 mm = very poorly.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 79 | 12 | 69 | 17
mm
  Baseline (n=70,0,68,0,71,74,75,79,0,69,0) | 62.47 (24.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 58.91 (22.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 54.62 (23.71) | 58.35 (23.14) | 56.09 (21.42) | 57.24 (25.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 51.88 (26.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=68,0,68,0,68,73,73,79,0,66,0) | 53.19 (22.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.96 (23.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.56 (22.89) | 42.32 (21.98) | 35.73 (21.46) | 41.80 (26.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.33 (25.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,65,0,67,70,72,76,0,66,0) | 47.87 (23.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.78 (22.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.94 (22.27) | 38.53 (24.49) | 34.76 (21.33) | 37.47 (25.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.21 (24.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,65,0,69,71,72,74,0,61,0) | 42.30 (22.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.08 (23.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.01 (24.06) | 35.41 (22.68) | 30.56 (21.87) | 34.86 (25.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.02 (25.14) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,62,0,66,67,70,73,0,61,0) | 41.06 (21.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.11 (22.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.50 (25.29) | 36.09 (24.38) | 30.61 (21.60) | 31.85 (25.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.64 (25.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=64,0,59,0,64,65,66,70,0,60,0) | 38.78 (22.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.42 (25.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 29.66 (21.69) | 35.05 (24.65) | 32.53 (24.48) | 30.76 (25.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.85 (25.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,45,13,58,66,61,54,12,37,16) | 30.76 (20.40) | 38.29 (19.76) | 29.84 (24.12) | 39.31 (27.48) | 30.62 (22.56) | 30.98 (22.06) | 26.59 (20.19) | 24.76 (22.53) | 50.67 (23.10) | 28.46 (22.69) | 37.63 (23.11)
  Week 20 (n=39,21,43,13,57,66,59,55,12,37,17) | 29.85 (22.86) | 37.95 (23.62) | 28.16 (22.36) | 42.08 (27.48) | 26.07 (22.75) | 35.00 (23.51) | 24.90 (20.57) | 25.56 (23.20) | 44.42 (27.38) | 26.22 (21.09) | 36.94 (27.13)
  Week 24 (n=40,20,44,13,55,64,60,53,12,36,17) | 28.23 (21.42) | 38.55 (27.08) | 25.93 (22.22) | 38.23 (27.28) | 23.64 (21.82) | 29.66 (21.58) | 25.07 (23.20) | 21.85 (18.07) | 34.83 (27.04) | 28.25 (21.49) | 34.59 (27.87)

13. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA) of Arthritis at Week 2, 4, 6, 8, 12, 16, 20 and 24/ET
Description: as for outcome 12
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 68 | 21 | 68 | 13 | 68 | 73 | 73 | 78 | 12 | 66 | 17
mm
  Week 2 (n=68,0,68,0,68,73,73,78,0,66,0) | -8.57 (26.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.96 (20.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -12.37 (21.83) | -16.74 (24.15) | -20.25 (26.92) | -15.38 (30.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.82 (24.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,65,0,67,70,72,75,0,66,0) | -13.90 (25.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -19.40 (25.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -15.70 (22.92) | -20.76 (26.76) | -21.82 (28.55) | -19.04 (29.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.65 (27.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,65,0,69,71,72,73,0,61,0) | -18.71 (29.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -22.02 (25.83) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -20.81 (24.06) | -24.03 (23.89) | -25.26 (30.85) | -22.99 (29.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.46 (23.90) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,62,0,66,67,70,72,0,61,0) | -20.35 (27.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -27.48 (26.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -17.44 (28.12) | -22.58 (25.37) | -24.81 (31.07) | -25.92 (30.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.48 (25.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=64,0,59,0,64,65,66,69,0,60,0) | -22.78 (28.81) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -23.95 (29.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -24.30 (24.57) | -24.77 (26.21) | -23.08 (30.87) | -28.09 (30.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -12.75 (28.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,45,13,58,66,61,53,12,37,16) | -33.60 (31.45) | -15.86 (22.28) | -28.00 (28.15) | -22.00 (26.01) | -24.05 (28.00) | -27.97 (24.02) | -28.90 (29.36) | -29.68 (31.20) | -13.67 (35.93) | -20.97 (31.57) | -14.81 (17.72)
  Week 20 (n=39,21,43,13,57,66,59,54,12,36,17) | -34.56 (31.99) | -16.19 (24.18) | -30.93 (25.67) | -19.23 (28.78) | -28.33 (26.93) | -23.95 (27.82) | -31.12 (32.09) | -30.67 (31.38) | -19.92 (34.52) | -23.22 (27.31) | -13.53 (22.22)
  Week 24 (n=40,20,44,13,55,64,60,53,12,36,17) | -36.68 (29.89) | -15.30 (32.99) | -32.11 (25.76) | -23.08 (31.06) | -29.84 (27.59) | -28.61 (25.31) | -30.83 (32.96) | -33.04 (32.02) | -29.50 (32.33) | -21.92 (27.51) | -15.88 (25.95)

14. Secondary Outcome: Physician Global Assessment of Arthritis
Description: Physician global assessment of arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 80 | 12 | 69 | 17
mm
  Baseline (n=70,0,68,0,71,74,75,80,0,69,0) | 62.66 (16.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 57.50 (18.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 56.51 (19.00) | 60.77 (16.75) | 60.51 (14.26) | 58.75 (17.90) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 58.30 (15.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=67,0,68,0,68,73,73,79,0,66,0) | 49.49 (21.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.07 (19.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.29 (20.12) | 42.85 (19.42) | 35.99 (15.97) | 41.92 (22.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 49.05 (18.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,65,0,67,70,72,75,0,66,0) | 41.69 (21.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.92 (21.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.73 (17.40) | 33.56 (19.77) | 33.35 (19.24) | 32.96 (22.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.23 (19.43) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,65,0,69,71,72,74,0,62,0) | 37.38 (17.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.51 (21.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 27.78 (18.40) | 30.82 (19.95) | 27.08 (17.28) | 32.65 (23.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.85 (21.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,62,0,66,67,70,73,0,61,0) | 35.71 (21.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 26.60 (20.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 27.26 (19.97) | 28.01 (19.90) | 23.06 (17.18) | 27.70 (21.09) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.66 (21.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=63,0,59,0,64,66,65,70,0,61,0) | 33.65 (20.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 26.17 (21.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 24.77 (18.80) | 26.47 (19.69) | 23.28 (17.89) | 28.93 (23.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.70 (24.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,44,13,58,66,61,55,12,37,16) | 23.95 (16.25) | 44.19 (24.68) | 19.77 (19.74) | 33.31 (22.97) | 23.67 (21.04) | 23.00 (18.60) | 19.31 (15.80) | 18.60 (15.00) | 48.42 (30.00) | 26.22 (18.43) | 27.44 (16.36)
  Week 20 (n=39,21,44,13,57,66,59,55,12,37,17) | 20.44 (18.10) | 34.29 (16.64) | 20.91 (18.21) | 32.92 (25.15) | 20.65 (18.68) | 24.05 (18.32) | 16.19 (12.41) | 18.84 (18.42) | 44.67 (25.31) | 21.95 (18.03) | 33.94 (22.43)
  Week 24 (n=40,19,43,13,55,64,60,53,11,36,17) | 18.90 (16.51) | 36.53 (21.17) | 20.26 (18.12) | 32.54 (24.26) | 16.91 (14.67) | 21.25 (17.79) | 14.68 (13.07) | 14.49 (11.75) | 41.00 (31.58) | 20.67 (15.81) | 32.18 (19.03)

15. Secondary Outcome: Change From Baseline in Physician Global Assessment of Arthritis at Week 2, 4, 6, 8, 12, 16, 20 and 24/ET
Description: as for outcome 14
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 67 | 21 | 68 | 13 | 68 | 73 | 73 | 79 | 12 | 68 | 17
mm
  Week 2 (n=67,0,68,0,68,73,73,79,0,66,0) | -12.88 (17.84) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -16.43 (19.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -14.60 (24.01) | -17.88 (17.66) | -24.30 (18.32) | -16.61 (19.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.82 (13.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,65,0,67,70,72,75,0,66,0) | -20.66 (19.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -20.80 (22.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -22.00 (20.79) | -27.67 (20.61) | -27.43 (21.04) | -25.31 (22.01) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -17.79 (18.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,65,0,69,71,72,74,0,62,0) | -25.02 (20.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -26.34 (24.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -28.80 (20.44) | -30.39 (20.61) | -33.26 (19.40) | -25.93 (23.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -20.15 (22.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,62,0,66,67,70,73,0,61,0) | -26.50 (22.83) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -30.92 (22.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -29.67 (24.30) | -33.63 (21.96) | -37.26 (19.37) | -30.66 (21.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -22.82 (22.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=63,0,59,0,64,66,66,70,0,61,0) | -28.76 (23.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -31.69 (24.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -31.58 (23.09) | -34.98 (20.53) | -36.80 (20.78) | -30.27 (22.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -21.77 (24.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,44,13,58,66,61,55,12,37,16) | -39.33 (19.85) | -16.95 (26.42) | -39.23 (23.11) | -23.85 (19.42) | -33.47 (26.06) | -38.45 (20.53) | -39.70 (20.34) | -38.65 (17.68) | -19.08 (29.20) | -29.89 (22.16) | -32.56 (15.65)
  Week 20 (n=39,21,44,13,57,66,59,55,12,37,17) | -42.21 (23.73) | -26.86 (23.81) | -38.70 (20.41) | -24.23 (22.29) | -36.81 (24.26) | -37.41 (18.99) | -43.42 (16.85) | -38.16 (19.33) | -22.83 (26.51) | -34.16 (23.25) | -26.29 (24.43)
  Week 24 (n=40,19,43,13,55,64,60,53,11,36,17) | -44.15 (22.39) | -24.11 (24.91) | -39.98 (21.13) | -24.62 (19.99) | -39.51 (22.83) | -40.61 (20.10) | -44.65 (16.76) | -41.91 (17.09) | -28.64 (31.29) | -35.06 (21.26) | -28.06 (20.84)

16. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 66 | 13 | 71 | 74 | 75 | 80 | 12 | 69 | 17
units on a scale
  Baseline (n=70,0,66,0,71,74,75,80,0,69,0) | 1.58 (0.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.36 (0.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.44 (0.64) | 1.33 (0.60) | 1.41 (0.64) | 1.46 (0.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.20 (0.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=68,0,68,0,68,73,73,79,0,66,0) | 1.41 (0.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.14 (0.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.20 (0.58) | 1.16 (0.61) | 1.15 (0.67) | 1.23 (0.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.15 (0.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,65,0,67,70,72,75,0,66,0) | 1.32 (0.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.03 (0.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.13 (0.65) | 1.08 (0.64) | 1.12 (0.69) | 1.14 (0.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.14 (0.66) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,64,0,69,71,72,74,0,61,0) | 1.23 (0.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.96 (0.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.03 (0.61) | 1.02 (0.65) | 1.05 (0.69) | 1.05 (0.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.07 (0.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,62,0,66,67,70,71,0,61,0) | 1.22 (0.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.93 (0.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.06 (0.66) | 0.89 (0.67) | 0.98 (0.68) | 0.98 (0.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.05 (0.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=64,0,59,0,64,65,66,68,0,61,0) | 1.19 (0.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.92 (0.75) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.94 (0.65) | 0.95 (0.68) | 0.96 (0.69) | 0.90 (0.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.08 (0.74) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,45,13,58,66,61,55,12,37,16) | 1.05 (0.59) | 1.42 (0.64) | 0.82 (0.72) | 1.18 (0.77) | 0.92 (0.60) | 0.91 (0.68) | 0.97 (0.75) | 0.81 (0.67) | 1.36 (0.67) | 0.80 (0.64) | 1.05 (0.80)
  Week 20 (n=39,21,44,13,57,66,59,55,12,37,17) | 0.95 (0.58) | 1.33 (0.72) | 0.77 (0.68) | 1.13 (0.78) | 0.78 (0.57) | 0.84 (0.65) | 0.92 (0.72) | 0.75 (0.63) | 1.42 (0.62) | 0.73 (0.65) | 0.92 (0.75)
  Week 24 (n=40,20,44,13,54,63,59,53,12,36,17) | 0.99 (0.57) | 1.38 (0.74) | 0.85 (0.68) | 1.05 (0.84) | 0.78 (0.62) | 0.85 (0.66) | 0.88 (0.69) | 0.72 (0.61) | 1.34 (0.78) | 0.74 (0.66) | 0.95 (0.68)

17. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 2, 4, 6, 8, 12, 16, 20 and 24/ET
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Change = scores at observation minus score at Baseline, and total possible score ranged from -3 to 3. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 68 | 21 | 66 | 13 | 68 | 73 | 73 | 79 | 12 | 66 | 17
units on a scale
  Week 2 (n=68,0,68,0,68,73,73,79,0,66,0) | -0.15 (0.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.23 (0.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.23 (0.41) | -0.18 (0.42) | -0.24 (0.40) | -0.23 (0.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.05 (0.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=68,0,63,0,67,70,72,75,0,66,0) | -0.24 (0.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.36 (0.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.32 (0.51) | -0.25 (0.45) | -0.31 (0.44) | -0.34 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.05 (0.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=66,0,62,0,69,71,72,74,0,61,0) | -0.31 (0.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.39 (0.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.42 (0.54) | -0.32 (0.57) | -0.34 (0.47) | -0.42 (0.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.13 (0.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=66,0,61,0,66,67,70,71,0,61,0) | -0.34 (0.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.41 (0.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.40 (0.58) | -0.43 (0.66) | -0.39 (0.49) | -0.50 (0.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.12 (0.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=64,0,58,0,64,65,66,68,0,61,0) | -0.37 (0.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.48 (0.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.51 (0.61) | -0.37 (0.63) | -0.45 (0.50) | -0.58 (0.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.10 (0.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,44,13,58,66,61,55,12,37,16) | -0.52 (0.48) | -0.16 (0.50) | -0.59 (0.64) | -0.08 (0.31) | -0.52 (0.59) | -0.41 (0.63) | -0.45 (0.60) | -0.62 (0.62) | -0.46 (0.58) | -0.30 (0.52) | -0.01 (0.29)
  Week 20 (n=39,21,43,13,57,66,59,55,12,37,17) | -0.62 (0.47) | -0.24 (0.42) | -0.62 (0.68) | -0.13 (0.41) | -0.64 (0.62) | -0.49 (0.58) | -0.51 (0.59) | -0.67 (0.65) | -0.41 (0.55) | -0.38 (0.54) | -0.11 (0.30)
  Week 24 (n=40,20,42,13,54,63,59,53,12,36,17) | -0.60 (0.52) | -0.21 (0.58) | -0.53 (0.65) | -0.21 (0.32) | -0.61 (0.65) | -0.47 (0.62) | -0.53 (0.60) | -0.66 (0.72) | -0.48 (0.74) | -0.37 (0.54) | -0.08 (0.29)

18. Secondary Outcome: C-Reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range of CRP is 0 milligram per deciliter (mg/dL) to 10 mg/dL. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 80 | 12 | 69 | 17
mg/dL
  Baseline (n=70,0,68,0,71,74,75,80,0,69,0) | 16.30 (18.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.85 (19.34) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 18.03 (24.96) | 14.42 (17.81) | 17.21 (16.94) | 14.68 (17.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 18.88 (19.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=65,0,63,0,63,69,68,74,0,61,0) | 14.54 (19.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.20 (11.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.98 (10.05) | 5.24 (9.59) | 4.08 (4.79) | 8.35 (13.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 18.10 (20.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=65,0,61,0,62,64,65,70,0,61,0) | 10.28 (11.83) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 10.11 (15.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.63 (12.54) | 5.46 (9.76) | 4.63 (8.68) | 8.67 (13.62) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.30 (16.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=64,0,61,0,66,67,66,69,0,58,0) | 10.55 (9.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.34 (13.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.26 (14.30) | 5.42 (10.04) | 5.41 (8.63) | 10.68 (17.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 15.18 (19.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=63,0,59,0,62,62,67,67,0,58,0) | 9.62 (11.78) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.64 (11.54) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.17 (11.47) | 10.18 (24.04) | 8.39 (11.39) | 9.75 (18.92) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 20.38 (30.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=61,0,57,0,60,63,62,65,0,60,0) | 8.53 (9.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.54 (13.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.54 (9.68) | 9.11 (20.08) | 5.81 (7.25) | 9.53 (15.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 19.69 (20.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,43,13,54,64,58,55,9,37,16) | 7.80 (10.30) | 7.02 (8.51) | 10.72 (18.93) | 5.85 (5.47) | 5.40 (8.06) | 6.77 (10.27) | 9.79 (22.24) | 6.52 (11.33) | 6.89 (7.06) | 13.08 (11.49) | 6.52 (7.30)
  Week 20 (n=39,21,44,13,57,63,57,55,12,36,17) | 8.96 (11.64) | 8.55 (12.87) | 7.71 (10.88) | 11.28 (17.83) | 7.93 (19.22) | 5.58 (8.69) | 3.46 (3.17) | 4.75 (5.28) | 7.89 (9.08) | 16.14 (16.63) | 12.10 (18.21)
  Week 24 (n=39,20,43,13,53,63,56,52,12,36,17) | 7.63 (10.26) | 6.02 (7.31) | 10.31 (17.43) | 12.58 (12.19) | 5.92 (14.78) | 6.66 (17.03) | 6.51 (11.04) | 4.54 (4.69) | 7.19 (8.18) | 13.39 (15.05) | 16.21 (26.51)

19. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 2, 4, 6, 8, 12, 16, 20 and 24/ET
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultra-sensitive assay. Normal range of CRP is 0 mg/dL to 10 mg/dL. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 65 | 21 | 63 | 13 | 63 | 69 | 68 | 74 | 12 | 61 | 17
mg/dL
  Week 2 (n=65,0,63,0,63,69,68,74,0,61,0) | -2.05 (18.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.93 (14.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.38 (19.27) | -9.19 (19.90) | -11.87 (15.22) | -6.56 (12.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.64 (14.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=65,0,61,0,62,64,65,70,0,61,0) | -6.07 (14.44) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.12 (17.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -8.54 (16.65) | -9.45 (16.27) | -11.70 (17.89) | -6.69 (13.99) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.26 (12.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=64,0,61,0,66,67,66,69,0,58,0) | -5.92 (16.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.97 (17.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.81 (23.67) | -9.38 (16.02) | -10.73 (17.63) | -5.03 (17.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.51 (12.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=63,0,59,0,62,62,67,67,0,58,0) | -5.94 (16.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.42 (14.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.35 (21.25) | -4.97 (24.54) | -8.67 (18.05) | -6.11 (19.97) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.70 (25.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=61,0,57,0,60,63,62,65,0,60,0) | -7.56 (17.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.28 (14.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -12.52 (23.93) | -5.96 (23.26) | -10.18 (16.26) | -5.71 (20.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.07 (15.90) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,43,13,54,64,58,55,9,37,16) | -6.96 (10.61) | -11.26 (21.64) | -7.04 (21.18) | -6.33 (10.48) | -11.53 (22.00) | -8.18 (18.99) | -7.01 (27.54) | -8.16 (17.01) | -7.59 (12.45) | -2.59 (13.79) | -13.44 (12.75)
  Week 20 (n=39,21,44,13,57,63,57,55,12,36,17) | -6.21 (10.94) | -9.73 (22.12) | -11.31 (16.46) | -0.90 (20.08) | -7.80 (23.28) | -9.60 (19.16) | -14.21 (16.73) | -9.65 (15.32) | -10.22 (13.83) | 0.11 (15.15) | -7.52 (20.34)
  Week 24 (n=39,20,43,43,53,63,56,52,12,36,17) | -7.61 (11.78) | -8.07 (10.28) | -7.57 (22.26) | 0.40 (16.50) | -8.18 (19.26) | -8.72 (22.73) | -10.65 (18.76) | -8.75 (15.40) | -10.92 (15.78) | -2.16 (16.06) | -3.41 (26.61)

20. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP])
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) less than or equal to (<=) 3.2 implied low disease activity and more than (>) 3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) less than (<) 2.6 = remission.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 80 | 12 | 69 | 17
units on a scale
  Baseline (n=70,0,68,0,71,74,75,79,0,69,0) | 5.48 (0.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.31 (0.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.14 (0.84) | 5.28 (0.85) | 5.39 (0.89) | 5.34 (0.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.26 (0.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=64,0,63,0,63,69,68,74,0,61,0) | 4.88 (1.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.46 (1.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.26 (0.90) | 4.18 (1.04) | 4.18 (1.16) | 4.28 (1.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.91 (1.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=65,0,61,0,62,64,65,70,0,61,0) | 4.45 (1.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.03 (1.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.03 (0.96) | 3.66 (1.12) | 3.75 (1.13) | 3.99 (1.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.60 (1.01) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=63,0,61,0,66,67,66,69,0,58,0) | 4.32 (1.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.74 (1.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.68 (1.00) | 3.59 (1.27) | 3.60 (1.13) | 3.94 (1.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.35 (1.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=63,0,59,0,62,62,67,67,0,58,0) | 4.21 (1.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.63 (1.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.54 (1.01) | 3.61 (1.23) | 3.38 (1.10) | 3.72 (1.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.30 (1.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=61,0,55,0,60,63,62,65,0,60,0) | 3.98 (1.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.46 (1.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.57 (1.09) | 3.40 (1.27) | 3.28 (1.25) | 3.61 (1.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.37 (1.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,43,13,54,64,58,55,9,37,16) | 3.59 (1.15) | 4.33 (1.16) | 3.11 (1.23) | 4.19 (1.48) | 3.19 (1.10) | 3.34 (1.22) | 3.12 (1.25) | 3.14 (1.06) | 4.65 (1.08) | 3.93 (1.06) | 3.91 (1.19)
  Week 20 (n=39,21,44,13,57,63,57,55,12,36,17) | 3.48 (1.28) | 3.83 (1.62) | 3.06 (1.25) | 4.24 (1.56) | 3.09 (1.17) | 3.14 (1.29) | 2.94 (1.04) | 3.08 (1.11) | 4.82 (1.24) | 3.81 (1.23) | 3.86 (1.24)
  Week 24 (n=39,20,42,13,53,63,56,52,12,36,17) | 3.39 (1.15) | 3.88 (1.49) | 3.14 (1.26) | 4.08 (1.35) | 3.03 (1.05) | 3.15 (1.19) | 2.91 (1.12) | 3.07 (0.98) | 4.51 (1.61) | 3.48 (1.06) | 4.08 (1.37)

21. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Week 2, 4, 6, 8, 12, 16, 20 and 24/ET
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 64 | 21 | 63 | 13 | 63 | 69 | 68 | 73 | 12 | 61 | 17
units on a scale
  Week 2 (n=64,0,63,0,63,69,68,73,0,61,0) | -0.55 (0.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.78 (0.92) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.86 (0.82) | -1.07 (0.84) | -1.22 (1.08) | -1.01 (0.97) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.26 (0.78) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=65,0,61,0,62,64,65,69,0,61,0) | -0.99 (0.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.23 (1.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.09 (0.94) | -1.58 (1.09) | -1.71 (1.20) | -1.30 (1.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.57 (0.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=63,0,61,0,66,67,66,69,0,58,0) | -1.13 (1.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.52 (1.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.44 (0.99) | -1.66 (1.18) | -1.81 (1.17) | -1.38 (1.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.80 (0.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=63,0,59,0,62,62,67,67,0,58,0) | -1.22 (1.14) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.61 (1.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.56 (0.97) | -1.63 (1.25) | -2.02 (1.14) | -1.63 (1.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.83 (1.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=61,0,55,0,60,63,62,65,0,60,0) | -1.45 (1.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.85 (1.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.59 (1.18) | -1.82 (1.17) | -2.13 (1.32) | -1.72 (1.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.82 (1.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,43,13,54,64,58,55,9,37,16) | -1.87 (1.13) | -1.14 (0.99) | -2.27 (1.14) | -0.81 (1.20) | -1.93 (1.12) | -1.89 (1.13) | -2.31 (1.39) | -2.13 (1.04) | -0.88 (0.95) | -1.14 (1.03) | -1.43 (0.70)
  Week 20 (n=39,21,44,13,57,63,57,55,12,36,17) | -1.94 (1.26) | -1.64 (1.25) | -2.41 (1.26) | -0.76 (1.22) | -2.05 (1.15) | -2.09 (1.28) | -2.49 (1.26) | -2.17 (0.96) | -0.95 (0.81) | -1.27 (1.37) | -1.47 (1.04)
  Week 24 (n=39,20,42,13,53,63,56,52,12,36,17) | -2.06 (1.22) | -1.55 (1.07) | -2.29 (1.19) | -0.92 (1.17) | -2.06 (1.04) | -2.13 (1.12) | -2.49 (1.27) | -2.19 (1.04) | -1.26 (1.23) | -1.55 (1.25) | -1.25 (0.96)

22. Secondary Outcome: Percentage of Participants With Categorization of Disease Improvement Based on DAS28-3 (CRP)
Description: Disease improvement was classified as good, moderate, and none based on improvement in DAS 28-3 (CRP) from baseline and present DAS 28-3 (CRP) score. Good: an improvement from baseline of >1.2 and a present score of <=3.2; none: an improvement of <=0.6 or >0.6 to <=1.2 with a present score of >5.1; remaining participants were classified as having moderate (Mod) improvement. Scores of good and moderate were considered to have therapeutic response.
Time Frame: Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 64 | 21 | 63 | 13 | 63 | 69 | 68 | 74 | 12 | 61 | 17
percentage of participants
  Week 2: Good (n=64,0,63,0,63,69,68,74,0,61,0) | 4.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 9.5 | 13.0 | 16.2 | 12.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.3 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Mod (n=64,0,63,0,63,69,68,74,0,61,0) | 23.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.9 | 46.4 | 50.0 | 41.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 23.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: None (n=64,0,63,0,63,69,68,74,0,61,0) | 71.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 50.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 47.6 | 40.6 | 33.8 | 44.6 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 73.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4: Good (n=65,0,61,0,62,64,65,70,0,61,0) | 10.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 21.3 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.1 | 28.1 | 30.8 | 21.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4: Mod (n=65,0,61,0,62,64,65,70,0,61,0) | 41.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 48.4 | 53.1 | 49.2 | 42.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4: None (n=65,0,61,0,62,64,65,70,0,61,0) | 47.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.5 | 18.8 | 20.0 | 34.3 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 57.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6: Good (n=63,0,61,0,66,67,66,69,0,58,0) | 11.1 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 29.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.8 | 29.9 | 31.8 | 23.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 12.1 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6: Mod (n=63,0,61,0,66,67,66,69,0,58,0) | 50.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.6 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.4 | 50.7 | 50.0 | 44.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.1 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6: None (n=63,0,61,0,66,67,66,69,0,58,0) | 38.1 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 27.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 25.8 | 19.4 | 18.2 | 31.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8: Good (n=63,0,59,0,62,62,67,67,0,58,0) | 19.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.1 | 32.3 | 43.3 | 37.3 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8: Mod (n=63,0,59,0,62,62,67,67,0,58,0) | 46.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 47.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.8 | 45.2 | 47.8 | 40.3 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.6 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8: None (n=63,0,59,0,62,62,67,67,0,58,0) | 34.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 22.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.1 | 22.6 | 9.0 | 22.4 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Good (n=61,0,55,0,60,63,62,65,0,60,0) | 23.0 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.3 | 41.3 | 51.6 | 36.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Mod (n=61,0,55,0,60,63,62,65,0,60,0) | 49.2 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 50.0 | 39.7 | 37.1 | 44.6 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: None (n=61,0,55,0,60,63,62,65,0,60,0) | 27.9 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 21.8 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.7 | 19.0 | 11.3 | 18.5 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.7 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16: Good (n=42,21,43,13,54,64,58,55,9,37,16) | 40.5 | 19.0 | 55.8 | 30.8 | 51.9 | 50.0 | 48.3 | 52.7 | 11.1 | 27.0 | 18.8
  Week 16: Mod (n=42,21,43,13,54,64,58,55,9,37,16) | 50.0 | 38.1 | 32.6 | 23.1 | 37.0 | 34.4 | 43.1 | 43.6 | 33.3 | 40.5 | 62.5
  Week 16: None (n=42,21,43,13,54,64,58,55,9,37,16) | 9.5 | 42.9 | 11.6 | 46.2 | 11.1 | 15.6 | 8.6 | 3.6 | 55.6 | 32.4 | 18.8
  Week 20: Good (n=39,21,44,13,57,63,57,55,12,36,17) | 46.2 | 42.9 | 59.1 | 15.4 | 61.4 | 52.4 | 57.9 | 52.7 | 0.0 | 30.6 | 29.4
  Week 20: Mod (n=39,21,44,13,57,63,57,55,12,36,17) | 43.6 | 28.6 | 31.8 | 46.2 | 28.1 | 36.5 | 35.1 | 40.0 | 58.3 | 36.1 | 47.1
  Week 20: None (n=39,21,44,13,57,63,57,55,12,36,17) | 10.3 | 28.6 | 9.1 | 38.5 | 10.5 | 11.1 | 7.0 | 7.3 | 41.7 | 33.3 | 23.5
  Week 24: Good (n=39,20,42,13,53,63,56,52,12,36,17) | 43.6 | 35.0 | 54.8 | 23.1 | 52.8 | 58.7 | 66.1 | 59.6 | 25.0 | 33.3 | 23.5
  Week 24: Mod (n=39,20,42,13,53,63,56,52,12,36,17) | 46.2 | 35.0 | 33.3 | 38.5 | 37.7 | 30.2 | 23.2 | 34.6 | 33.3 | 41.7 | 47.1
  Week 24: None (n=39,20,42,13,53,63,56,52,12,36,17) | 10.3 | 30.0 | 11.9 | 38.5 | 9.4 | 11.1 | 10.7 | 5.8 | 41.7 | 25.0 | 29.4

23. Secondary Outcome: Percentage of Participants With Disease Remission Based on DAS28-3 (CRP)
Description: DAS28-3 (CRP) defined remission was classified as a score of <2.6.
Time Frame: Week 2, 4, 6, 8, 12, 16, 20, 24/ET
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 64 | 21 | 63 | 13 | 63 | 68 | 68 | 74 | 12 | 61 | 17
percentage of participants
  Week 2 (n=64,0,63,0,63,68,68,74,0,61,0) | 1.56 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.17 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.59 | 4.41 | 13.24 | 4.05 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.28 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 4 (n=65,0,61,0,62,63,65,70,0,61,0) | 4.62 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 14.75 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.06 | 19.05 | 16.92 | 10.00 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.28 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 6 (n=63,0,61,0,66,66,66,69,0,58,0) | 3.17 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 19.67 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.64 | 24.24 | 22.73 | 10.14 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.45 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 8 (n=63,0,59,0,62,61,67,67,0,58,0) | 7.94 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 22.03 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 19.35 | 21.31 | 23.88 | 20.90 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.90 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=61,0,55,0,60,62,62,65,0,60,0) | 6.56 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.91 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 16.67 | 32.26 | 37.10 | 24.62 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.67 | NA — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 16 (n=42,21,43,13,54,63,58,55,9,37,16) | 14.3 | 9.5 | 41.9 | 23.1 | 24.1 | 30.2 | 37.9 | 29.1 | 11.1 | 8.1 | 12.5
  Week 20 (n=39,21,44,13,57,62,57,55,12,36,17) | 20.5 | 28.6 | 43.2 | 15.4 | 35.1 | 37.1 | 38.6 | 30.9 | 0.0 | 13.9 | 17.6
  Week 24 (n=39,20,42,13,53,63,56,52,12,36,17) | 23.1 | 25.0 | 35.7 | 15.4 | 41.5 | 36.5 | 39.3 | 32.7 | 16.7 | 19.4 | 17.6

24. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36)
Description: SF-36 is a standardized survey evaluating 8 domains (of 2 components [C]; physical [Ph] and mental [Mn]) of functional health and well being: physical and social (So) functioning (Fn), physical and emotional role (role-physical [R-P], role-emotional [R-E]) limitations, bodily pain (BP), general health (GH), vitality (Vit), mental health (MnH). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline, Week 12, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 20 | 68 | 13 | 71 | 73 | 75 | 80 | 12 | 69 | 17
units on a scale
  Baseline: Ph Fn (n=70,0,68,0,71,73,75,80,0,69,0) | 31.48 (10.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.20 (11.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.93 (9.66) | 31.92 (9.15) | 31.50 (9.29) | 30.23 (9.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.01 (11.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: R-P (n=70,0,68,0,71,73,75,80,0,69,0) | 34.53 (8.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.45 (10.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.54 (8.69) | 34.64 (10.72) | 33.70 (9.85) | 33.13 (9.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.23 (9.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: BP (n=70,0,68,0,71,73,75,80,0,69,0) | 34.14 (6.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.60 (8.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.36 (8.23) | 35.11 (7.85) | 34.98 (8.19) | 34.20 (8.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.93 (8.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: GH (n=70,0,68,0,71,73,75,80,0,69,0) | 35.08 (6.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.17 (8.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.12 (8.90) | 36.52 (9.28) | 35.94 (8.44) | 36.08 (8.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.50 (9.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Vit (n=70,0,68,0,71,73,75,80,0,69,0) | 40.32 (9.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.36 (10.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.54 (9.39) | 42.60 (10.83) | 40.81 (11.75) | 40.97 (9.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.08 (11.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: So Fn (n=70,0,68,0,71,73,75,80,0,69,0) | 37.76 (10.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.88 (11.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.72 (10.38) | 38.99 (10.80) | 38.01 (11.06) | 38.03 (10.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.09 (11.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: R-E (n=70,0,68,0,71,73,75,80,0,69,0) | 34.72 (11.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.18 (14.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.21 (12.51) | 36.23 (12.64) | 34.73 (14.42) | 35.13 (13.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.37 (13.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: MnH (n=70,0,68,0,71,73,75,80,0,69,0) | 38.98 (11.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.07 (11.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.88 (12.02) | 42.79 (10.99) | 39.68 (12.65) | 39.91 (12.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.91 (13.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Ph C (n=70,0,68,0,71,73,75,80,0,69,0) | 33.13 (6.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.73 (8.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.99 (8.03) | 32.96 (8.15) | 33.19 (7.31) | 32.11 (8.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.41 (8.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Mn C (n=70,0,68,0,71,73,75,80,0,69,0) | 40.39 (11.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.47 (12.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.81 (11.80) | 43.53 (11.00) | 40.92 (13.00) | 41.68 (12.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.72 (13.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Ph Fn (n=63,0,59,0,64,65,65,70,0,61,0) | 35.05 (10.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.49 (11.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.45 (9.78) | 36.25 (10.75) | 37.80 (10.76) | 37.49 (11.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 36.23 (11.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: R-P (n=63,0,59,0,64,65,65,70,0,61,0) | 38.47 (8.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.25 (10.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.26 (10.21) | 39.71 (9.69) | 39.41 (10.03) | 40.17 (10.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.79 (10.14) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: BP (n=63,0,59,0,64,65,65,70,0,61,0) | 41.62 (8.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.76 (11.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.73 (9.57) | 44.00 (10.81) | 44.39 (9.40) | 44.21 (9.78) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.46 (10.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: GH (n=63,0,59,0,64,65,65,70,0,61,0) | 37.85 (8.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.04 (8.74) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.11 (9.54) | 39.15 (8.76) | 40.05 (9.44) | 41.10 (9.78) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.54 (10.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Vit (n=63,0,59,0,64,65,65,70,0,61,0) | 45.45 (9.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.80 (10.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.33 (10.59) | 45.99 (10.68) | 47.82 (10.24) | 46.03 (11.42) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.48 (12.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: So Fn (n=63,0,59,0,64,65,65,70,0,61,0) | 41.18 (11.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.54 (11.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.28 (10.82) | 42.84 (10.06) | 43.93 (9.81) | 44.23 (10.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.38 (10.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: R-E (n=63,0,59,0,64,65,65,70,0,61,0) | 39.47 (12.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.14 (12.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.90 (12.87) | 39.01 (12.07) | 39.07 (11.96) | 41.33 (13.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.39 (12.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: MnH (n=63,0,59,0,64,65,65,70,0,61,0) | 43.84 (10.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.57 (10.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.34 (13.08) | 43.08 (9.84) | 45.24 (10.70) | 46.11 (11.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.36 (12.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Ph C (n=63,0,59,0,64,65,65,70,0,61,0) | 37.24 (8.19) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.70 (9.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.27 (9.31) | 39.52 (9.30) | 39.97 (8.98) | 39.64 (10.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.89 (9.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Mn C (n=63,0,59,0,64,65,65,70,0,61,0) | 44.86 (11.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.47 (11.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.84 (13.41) | 44.18 (10.26) | 45.61 (10.59) | 46.65 (11.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.08 (12.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24: Ph Fn(n=40,20,44,13,55,64,60,53,12,36,17) | 37.41 (10.35) | 34.30 (10.72) | 38.38 (11.35) | 39.39 (11.83) | 40.04 (10.81) | 38.19 (10.88) | 38.62 (11.08) | 40.51 (12.11) | 32.31 (11.36) | 39.44 (10.64) | 38.09 (10.04)
  Week 24: R-P (n=40,20,44,13,55,64,60,53,12,36,17) | 40.51 (8.53) | 35.06 (9.36) | 39.88 (11.85) | 38.96 (10.26) | 41.09 (9.12) | 40.32 (10.91) | 40.69 (9.67) | 41.97 (10.80) | 35.02 (10.72) | 44.27 (9.80) | 42.45 (9.44)
  Week 24: BP (n=40,20,44,13,55,64,60,53,12,36,17) | 44.17 (8.68) | 39.57 (11.54) | 44.15 (10.31) | 43.07 (9.91) | 44.96 (9.23) | 44.52 (10.98) | 45.76 (9.67) | 46.89 (10.25) | 40.32 (11.00) | 43.11 (9.54) | 44.24 (8.09)
  Week 24: GH (n=40,20,44,13,55,64,60,53,12,36,17) | 40.65 (7.40) | 36.87 (7.75) | 41.45 (10.05) | 37.35 (5.95) | 41.35 (10.23) | 41.09 (9.27) | 41.40 (9.24) | 44.03 (9.52) | 35.81 (11.52) | 43.16 (9.70) | 40.68 (8.34)
  Week 24: Vit (n=40,20,44,13,55,64,60,53,12,36,17) | 49.05 (10.69) | 39.60 (9.23) | 48.76 (11.25) | 47.29 (6.58) | 48.40 (10.41) | 47.55 (10.18) | 50.11 (11.68) | 50.50 (10.98) | 41.94 (13.65) | 49.75 (11.83) | 48.23 (11.92)
  Week 24: So Fn(n=40,20,44,13,55,64,60,53,12,36,17) | 43.62 (10.40) | 39.40 (10.26) | 42.84 (12.53) | 43.84 (9.05) | 45.25 (11.64) | 43.56 (10.73) | 44.67 (10.31) | 46.35 (10.53) | 38.67 (12.38) | 45.18 (10.60) | 43.05 (10.04)
  Week 24: R-E (n=40,20,44,13,55,64,60,53,12,36,17) | 40.23 (11.08) | 34.30 (10.59) | 40.59 (13.86) | 37.94 (12.35) | 41.46 (12.40) | 40.15 (11.58) | 40.39 (11.88) | 42.31 (13.71) | 37.09 (16.56) | 42.27 (13.09) | 46.28 (9.13)
  Week 24: MnH (n=40,20,44,13,55,64,60,53,12,36,17) | 45.92 (11.10) | 38.74 (10.58) | 45.66 (12.59) | 44.59 (7.04) | 47.29 (13.62) | 43.89 (10.93) | 46.86 (11.73) | 47.24 (11.36) | 43.44 (12.84) | 45.63 (14.22) | 47.52 (11.26)
  Week 24: Ph C (n=40,20,44,13,55,64,60,53,12,36,17) | 39.94 (8.41) | 36.79 (9.76) | 40.31 (9.95) | 39.74 (9.76) | 41.12 (9.22) | 40.85 (9.79) | 40.99 (9.14) | 42.81 (10.22) | 34.40 (10.57) | 42.09 (9.20) | 39.41 (9.58)
  Week 24: Mn C(n=40,20,44,13,55,64,60,53,12,36,17) | 46.62 (12.04) | 39.10 (11.18) | 46.21 (13.26) | 44.52 (7.18) | 47.34 (13.41) | 45.03 (11.20) | 47.21 (11.71) | 48.03 (11.81) | 43.35 (13.89) | 47.08 (15.31) | 49.27 (9.52)

25. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) at Week 12 and 24/ET
Description: as for outcome 24
Time Frame: Baseline, Week 12, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 63 | 20 | 59 | 13 | 64 | 64 | 65 | 70 | 12 | 61 | 17
units on a scale
  Week 12: Ph Fn (n=63,0,59,0,64,64,65,70,0,61,0) | 3.98 (7.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.39 (9.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.57 (8.25) | 4.18 (11.13) | 5.96 (8.21) | 7.40 (9.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.24 (8.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: R-P (n=63,0,59,0,64,64,65,70,0,61,0) | 3.77 (8.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.61 (11.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.68 (9.44) | 4.52 (11.62) | 5.20 (9.27) | 6.86 (9.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.01 (9.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: BP (n=63,0,59,0,64,64,65,70,0,61,0) | 7.29 (8.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.80 (11.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.28 (10.29) | 8.74 (10.66) | 9.23 (9.48) | 10.54 (9.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.23 (8.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: GH (n=63,0,59,0,64,64,65,70,0,61,0) | 2.94 (7.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.84 (7.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.78 (8.81) | 2.73 (7.46) | 4.32 (8.59) | 4.97 (9.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.47 (10.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Vit (n=63,0,59,0,64,64,65,70,0,61,0) | 5.10 (8.99) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.29 (9.92) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.68 (9.86) | 2.29 (8.80) | 6.87 (8.76) | 5.22 (8.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.45 (11.66) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: So Fn (n=63,0,59,0,64,64,65,70,0,61,0) | 3.72 (10.54) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.99 (10.54) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.26 (9.93) | 3.49 (11.84) | 4.70 (10.33) | 5.84 (12.43) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.80 (9.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: R-E (n=63,0,59,0,64,64,65,70,0,61,0) | 4.26 (10.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.69 (13.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.25 (11.23) | 2.73 (13.28) | 3.77 (13.04) | 5.33 (12.06) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.96 (12.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: MnH (n=63,0,59,0,64,64,65,70,0,61,0) | 4.92 (9.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.63 (10.01) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.43 (10.19) | 0.04 (9.08) | 4.68 (8.73) | 5.59 (9.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.88 (9.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Ph C (n=63,0,59,0,64,64,65,70,0,61,0) | 4.27 (6.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.16 (8.82) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.30 (8.03) | 6.32 (8.72) | 6.77 (7.29) | 7.98 (7.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.71 (7.43) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Mn C (n=63,0,59,0,64,64,65,70,0,61,0) | 4.30 (9.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.94 (10.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.72 (9.57) | 0.28 (10.13) | 3.81 (9.58) | 4.18 (10.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.40 (9.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24: Ph Fn(n=40,20,44,13,55,63,60,53,12,36,17) | 6.52 (8.32) | 2.63 (9.94) | 5.45 (8.57) | 4.37 (8.35) | 7.77 (9.41) | 6.41 (11.62) | 6.63 (10.30) | 8.81 (10.48) | 6.49 (8.15) | 3.74 (9.56) | 4.21 (9.84)
  Week 24: R-P (n=40,20,44,13,55,63,60,53,12,36,17) | 6.12 (8.34) | 1.47 (7.72) | 5.07 (11.00) | 4.52 (6.77) | 6.01 (10.23) | 5.56 (9.76) | 6.61 (9.33) | 7.25 (11.27) | 5.51 (10.50) | 5.85 (11.43) | 4.75 (8.64)
  Week 24: BP (n=40,20,44,13,55,63,60,53,12,36,17) | 10.65 (9.91) | 3.85 (8.92) | 10.16 (9.54) | 9.75 (7.27) | 10.09 (10.44) | 9.21 (10.31) | 10.44 (10.51) | 11.86 (10.67) | 10.67 (12.01) | 5.92 (10.51) | 7.73 (7.63)
  Week 24: GH (n=40,20,44,13,55,63,60,53,12,36,17) | 5.62 (7.70) | 3.58 (6.97) | 5.92 (7.09) | 4.11 (9.07) | 6.34 (7.85) | 4.68 (8.77) | 5.41 (7.88) | 6.43 (8.93) | 5.92 (9.84) | 4.20 (12.05) | 4.04 (3.82)
  Week 24: Vit (n=40,20,44,13,55,63,60,53,12,36,17) | 8.12 (9.94) | 1.56 (10.79) | 5.82 (9.30) | 5.04 (10.16) | 6.64 (9.03) | 3.52 (9.27) | 8.53 (9.99) | 7.95 (11.17) | 6.76 (11.52) | 2.08 (13.86) | 6.06 (6.19)
  Week 24: So Fn(n=40,20,44,13,55,63,60,53,12,36,17) | 5.86 (9.36) | 3.27 (12.31) | 4.09 (11.10) | 5.87 (10.31) | 7.54 (10.36) | 4.16 (11.99) | 4.91 (10.27) | 6.79 (11.86) | 3.64 (11.71) | 3.33 (12.73) | 3.85 (9.20)
  Week 24: R-E (n=40,20,44,13,55,63,60,53,12,36,17) | 4.28 (11.30) | 2.33 (12.82) | 5.48 (16.05) | -0.30 (13.69) | 4.24 (11.81) | 4.01 (13.30) | 5.18 (11.73) | 5.57 (14.61) | 2.27 (16.86) | 0.97 (13.70) | 2.29 (11.17)
  Week 24: MnH (n=40,20,44,13,55,63,60,53,12,36,17) | 7.25 (12.82) | 1.83 (8.73) | 4.99 (11.52) | 4.98 (11.27) | 5.43 (11.92) | 0.36 (10.48) | 5.44 (8.23) | 5.31 (12.73) | 6.57 (12.84) | 0.70 (9.97) | 0.99 (10.10)
  Week 24: Ph C (n=40,20,44,13,55,63,60,53,12,36,17) | 7.47 (7.90) | 2.91 (7.31) | 6.78 (7.17) | 6.62 (5.93) | 8.31 (8.48) | 7.99 (9.21) | 7.81 (8.84) | 9.59 (8.67) | 7.83 (7.89) | 6.26 (9.97) | 6.40 (8.08)
  Week 24: Mn C (n=40,20,44,13,55,63,60,53,12,36,17) | 5.48 (12.35) | 1.93 (11.99) | 4.31 (13.10) | 2.48 (11.80) | 4.46 (10.55) | 0.73 (10.85) | 4.78 (9.04) | 4.52 (12.52) | 3.44 (14.10) | -0.07 (12.42) | 1.57 (8.22)

26. Secondary Outcome: Euro Quality of Life-5 Dimentions (EQ-5D) - Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQoL Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Week 12, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 80 | 12 | 69 | 17
units on a scale
  Baseline (n=70,0,68,0,71,74,75,80,0,69,0) | 0.45 (0.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.46 (0.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.50 (0.30) | 0.48 (0.28) | 0.46 (0.31) | 0.49 (0.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.49 (0.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=63,0,59,0,64,65,64,70,0,61,0) | 0.63 (0.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.59 (0.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.62 (0.26) | 0.65 (0.23) | 0.63 (0.27) | 0.64 (0.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.55 (0.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24 (n=40,20,44,13,55,63,60,52,12,36,17) | 0.66 (0.23) | 0.46 (0.42) | 0.67 (0.26) | 0.64 (0.25) | 0.70 (0.23) | 0.68 (0.23) | 0.65 (0.25) | 0.71 (0.27) | 0.56 (0.32) | 0.65 (0.22) | 0.58 (0.32)

27. Secondary Outcome: Change From Baseline in Euro Quality of Life-5 Dimentions (EQ-5D) - Health State Profile Utility at Week 12 and 24/ET
Description: as for outcome 26
Time Frame: Baseline, Week 12, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 63 | 20 | 59 | 13 | 64 | 65 | 64 | 70 | 12 | 61 | 17
units on a scale
  Week 12 (n=63,0,59,0,64,65,64,70,0,61,0) | 0.15 (0.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.16 (0.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.11 (0.32) | 0.17 (0.27) | 0.18 (0.29) | 0.16 (0.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.05 (0.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24 (n=40,20,44,13,55,63,60,52,12,36,17) | 0.20 (0.30) | 0.00 (0.30) | 0.23 (0.33) | 0.23 (0.37) | 0.19 (0.30) | 0.20 (0.31) | 0.18 (0.29) | 0.17 (0.32) | 0.20 (0.45) | 0.13 (0.30) | 0.03 (0.29)

28. Secondary Outcome: Medical Outcome Study- Sleep Scale (MOS-SS)
Description: Participant-rated questionnaire to assess key constructs of sleep over the past week. Consists of a 12-item based on 7 subscales: sleep disturbance (SD), snoring (Sno), awakened short of breath (ASOB) or with headache, sleep adequacy (Ade), and somnolence (Som) (range:0-100); sleep quantity (Qua)(range:0-24), and optimal (Opt) sleep (yes: 1, no: 0)and nine item index measures of sleep disturbance were constructed to provide composite scores: sleep problem summary (SPS) and overall sleep problems (OSP). Except sleep adequacy, optimal sleep and quantity, higher scores=greater impairment. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range* 100); total score range: 0 to 100; higher score = greater intensity of attribute.
Time Frame: Baseline, Week 2, 12, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 74 | 75 | 80 | 12 | 69 | 17
units on a scale
  Baseline: SPS (n=70,0,68,0,71,74,74,80,0,69,0) | 40.62 (18.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.46 (21.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.12 (18.93) | 36.94 (18.49) | 40.90 (22.41) | 38.46 (21.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.26 (19.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: OSP (n=70,0,68,0,71,74,74,79,0,69,0) | 41.94 (18.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 45.65 (20.86) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.22 (19.00) | 39.05 (18.56) | 42.87 (20.62) | 40.49 (21.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.86 (19.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Ade (n=70,0,68,0,71,74,74,80,0,69,0) | 48.14 (25.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 43.82 (26.99) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 46.20 (27.95) | 50.27 (26.84) | 49.19 (28.13) | 51.00 (30.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 51.45 (28.45) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: ASOB (n=70,0,68,0,71,74,75,80,0,69,0) | 20.00 (24.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 22.94 (24.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.75 (22.82) | 17.30 (22.29) | 21.87 (25.93) | 20.50 (27.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 22.61 (25.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: SD (n=70,0,68,0,71,74,75,80,0,69,0) | 44.43 (23.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 49.10 (27.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 42.61 (25.40) | 41.17 (25.36) | 48.37 (25.66) | 44.42 (27.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 40.34 (26.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Opt (n=70,0,68,0,71,74,75,80,0,69,0) | 0.51 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.44 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.46 (0.50) | 0.45 (0.50) | 0.47 (0.50) | 0.50 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.52 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Qua (n=70,0,67,0,71,74,75,78,0,69,0) | 6.87 (1.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.72 (1.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.32 (7.65) | 7.28 (3.54) | 6.64 (1.61) | 6.90 (1.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.71 (1.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Sno (n=69,0,68,0,71,74,74,80,0,69,0) | 31.59 (30.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.29 (32.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 44.51 (33.16) | 39.73 (33.19) | 36.00 (34.01) | 35.25 (32.49) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.94 (33.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Baseline: Som (n=70,0,68,0,71,74,75,78,0,69,0) | 35.14 (20.30) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 38.63 (23.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.86 (19.17) | 34.50 (19.03) | 35.91 (22.08) | 35.04 (22.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.04 (20.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: SPS (n=67,0,68,0,68,73,73,79,0,65,0) | 39.65 (21.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.89 (22.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.22 (21.10) | 35.25 (19.10) | 32.97 (21.75) | 35.78 (20.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.34 (20.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: OSP (n=68,0,68,0,68,73,73,79,0,66,0) | 39.04 (19.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.88 (21.48) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.74 (20.11) | 35.65 (19.37) | 35.27 (20.56) | 36.22 (19.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.67 (18.79) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Ade (n=68,0,68,0,68,73,73,79,0,66,0) | 45.15 (27.62) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 49.56 (28.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 53.24 (31.64) | 53.42 (25.40) | 57.53 (28.81) | 50.51 (27.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 54.24 (29.87) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: ASOB (n=68,0,68,0,68,73,73,79,0,65,0) | 20.29 (25.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.65 (22.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.94 (22.70) | 22.74 (24.11) | 15.34 (21.74) | 20.25 (26.11) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 17.88 (23.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: SD (n=68,0,68,0,68,73,73,79,0,66,0) | 39.15 (22.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 39.21 (27.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.00 (23.80) | 34.93 (24.83) | 38.73 (26.23) | 35.87 (24.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.33 (25.29) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Opt (n=68,0,68,0,68,73,73,79,0,66,0) | 0.41 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.43 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.53 (0.50) | 0.52 (0.50) | 0.52 (0.50) | 0.44 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.59 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Qua (n=68,0,68,0,68,73,73,79,0,66,0) | 6.75 (1.73) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.76 (1.40) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.72 (1.26) | 7.05 (1.30) | 7.10 (1.70) | 6.78 (1.65) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.08 (1.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Sno (n=68,0,67,0,68,73,73,79,0,66,0) | 32.94 (29.88) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.59 (32.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 37.01 (31.38) | 35.62 (33.21) | 30.96 (33.01) | 30.63 (30.18) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.76 (35.17) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Som (n=67,0,68,0,68,73,73,79,0,66,0) | 32.34 (21.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.63 (24.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.08 (21.66) | 33.79 (20.97) | 32.69 (21.26) | 31.73 (22.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.51 (20.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: SPS (n=62,0,59,0,63,65,64,70,0,61,0) | 35.05 (16.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.62 (22.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.39 (20.64) | 34.92 (18.85) | 35.00 (19.41) | 32.81 (21.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.26 (22.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: OSP (n=62,0,59,0,63,65,64,70,0,61,0) | 34.78 (16.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.23 (20.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.61 (19.83) | 35.26 (19.48) | 36.33 (19.86) | 33.44 (21.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.50 (20.96) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Ade (n=62,0,59,0,63,65,64,70,0,61,0) | 49.35 (24.69) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 54.92 (32.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 53.17 (29.99) | 54.00 (26.74) | 56.09 (28.21) | 58.43 (27.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 54.59 (27.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: ASOB (n=62,0,59,0,63,65,64,70,0,61,0) | 15.16 (22.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 13.90 (19.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 20.32 (27.24) | 20.00 (23.72) | 18.75 (22.50) | 21.43 (26.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 20.98 (28.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: SD (n=62,0,59,0,63,65,64,70,0,61,0) | 34.94 (20.00) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.66 (26.03) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.52 (23.96) | 34.27 (25.00) | 39.16 (25.16) | 34.18 (27.10) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.41 (26.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Opt (n=63,0,59,0,64,65,65,70,0,61,0) | 0.52 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.53 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.48 (0.50) | 0.54 (0.50) | 0.45 (0.50) | 0.51 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.48 (0.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Qua (n=62,0,58,0,63,65,64,70,0,61,0) | 7.08 (1.41) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 7.05 (1.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.71 (1.49) | 6.85 (1.33) | 6.98 (1.74) | 7.60 (5.37) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 8.10 (9.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Sno (n=61,0,59,0,63,65,64,70,0,61,0) | 29.18 (26.97) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.92 (32.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 41.59 (32.19) | 35.69 (32.11) | 34.69 (32.71) | 33.43 (29.63) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 30.82 (31.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Som (n=62,0,59,0,63,65,64,70,0,61,0) | 28.82 (18.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.20 (21.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 31.01 (23.10) | 34.36 (23.22) | 32.29 (20.62) | 30.57 (25.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 28.96 (18.77) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24: SPS (n=40,20,44,13,55,64,59,52,12,34,17) | 32.17 (17.35) | 43.67 (20.23) | 30.68 (21.02) | 38.21 (17.46) | 32.55 (22.35) | 32.50 (18.22) | 29.89 (18.91) | 25.45 (17.75) | 44.44 (27.09) | 29.51 (19.04) | 32.55 (22.31)
  Week 24: OSP (n=40,20,44,13,55,64,59,52,12,34,17) | 31.64 (16.38) | 42.86 (19.06) | 31.46 (19.54) | 38.80 (18.07) | 32.18 (21.24) | 32.95 (18.88) | 31.18 (19.77) | 26.76 (17.75) | 47.27 (27.08) | 30.41 (18.52) | 33.04 (21.93)
  Week 24: Ade (n=40,20,44,13,55,64,59,52,12,34,17) | 57.00 (25.74) | 39.50 (27.81) | 58.41 (28.69) | 46.15 (18.05) | 55.64 (31.61) | 57.34 (26.32) | 57.46 (26.43) | 66.92 (28.60) | 44.17 (34.50) | 57.65 (27.64) | 55.29 (33.56)
  Week 24: ASOB (n=40,20,44,13,55,64,59,52,12,34,17 | 14.00 (17.66) | 20.00 (26.75) | 12.73 (18.85) | 18.46 (17.25) | 14.18 (20.61) | 17.19 (23.33) | 11.53 (19.72) | 11.15 (18.33) | 25.00 (32.05) | 13.53 (15.35) | 14.12 (25.26)
  Week 24: SD (n=40,20,44,13,55,64,59,52,12,34,17) | 32.31 (19.05) | 40.19 (21.76) | 30.80 (24.04) | 38.08 (28.62) | 32.77 (25.76) | 32.73 (26.78) | 32.61 (26.23) | 28.49 (23.70) | 52.19 (29.21) | 30.33 (24.00) | 36.40 (27.29)
  Week 24: Opt (n=40,20,44,13,55,64,60,53,12,36,17) | 0.53 (0.51) | 0.50 (0.51) | 0.55 (0.50) | 0.38 (0.51) | 0.45 (0.50) | 0.55 (0.50) | 0.45 (0.50) | 0.57 (0.50) | 0.33 (0.49) | 0.58 (0.50) | 0.41 (0.51)
  Week 24: Qua (n=40,20,44,13,55,64,59,52,12,34,17) | 6.88 (1.44) | 6.80 (1.40) | 7.25 (1.31) | 6.69 (1.65) | 7.93 (7.26) | 6.94 (1.23) | 7.05 (1.85) | 7.12 (1.20) | 9.42 (12.87) | 7.43 (1.09) | 6.41 (1.42)
  Week 24: Sno (n=40,20,44,13,54,64,59,52,12,34,17) | 26.50 (23.70) | 38.00 (32.38) | 35.00 (31.73) | 44.62 (32.82) | 37.41 (32.05) | 38.13 (33.37) | 35.25 (30.25) | 38.46 (32.62) | 35.00 (28.44) | 27.06 (32.62) | 34.12 (33.74)
  Week 24: Som (n=40,20,44,13,55,64,59,52,12,34,17) | 29.50 (19.33) | 40.67 (20.85) | 34.39 (25.39) | 31.79 (18.49) | 29.94 (20.68) | 32.40 (24.05) | 28.70 (19.93) | 26.03 (21.42) | 33.89 (25.34) | 27.06 (17.67) | 23.14 (18.12)

29. Secondary Outcome: Change From Baseline in Medical Outcome Study- Sleep Scale (MOS-SS) at Week 2, 12 and 24/ET
Description: Participant-rated questionnaire to assess key constructs of sleep over the past week. Consists of a 12-item based on 7 subscales: sleep disturbance (SD), snoring (Sno), awakened short of breath (ASOB) or with headache, sleep adequacy (Ade), and somnolence (Som) (range: 0-100); sleep quantity (Qua) (range: 0-24), and optimal (Opt) sleep (yes: 1, no: 0) and 9 item index measures of sleep disturbance were constructed to provide 2 composite scores: sleep problem summary (SPS) and overall sleep problems (OSP). Except sleep adequacy, optimal sleep and quantity, higher scores=greater impairment. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range*100); total score range: 0 to 100; higher score = greater intensity of attribute.
Time Frame: Baseline, Week 2, 12, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 67 | 20 | 68 | 13 | 68 | 73 | 72 | 79 | 12 | 66 | 17
units on a scale
  Week 2: SPS (n=67,0,68,0,68,73,72,79,0,66,0) | -0.95 (11.35) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.57 (15.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.43 (16.51) | -2.05 (14.11) | -7.45 (11.74) | -2.36 (17.85) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.29 (13.12) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: OSP (n=67,0,68,0,68,73,72,78,0,65,0) | -2.94 (10.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.76 (14.28) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.93 (14.92) | -3.75 (12.36) | -7.06 (10.93) | -4.07 (15.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.30 (12.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Ade (n=68,0,68,0,68,73,72,79,0,66,0) | -3.68 (22.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.74 (21.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 6.76 (25.06) | 3.70 (26.11) | 7.64 (16.74) | -0.51 (28.68) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.18 (19.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: ASOB (n=68,0,68,0,68,73,73,79,0,66,0) | -0.29 (19.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.29 (20.62) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.29 (25.27) | 5.48 (21.15) | -6.03 (21.78) | 0.00 (20.51) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.76 (25.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: SD (n=68,0,68,0,68,73,73,79,0,65,0) | -5.64 (13.23) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.89 (17.97) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.82 (18.04) | -6.73 (15.61) | -8.77 (15.11) | -7.85 (20.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.81 (17.05) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Opt (n=68,0,68,0,68,73,73,79,0,66,0) | -0.10 (0.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.01 (0.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.04 (0.44) | 0.07 (0.56) | 0.04 (0.54) | -0.05 (0.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.08 (0.36) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Qua (n=68,0,67,0,68,73,73,77,0,66,0) | -0.13 (1.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.03 (1.07) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.69 (7.75) | -0.21 (3.75) | 0.41 (1.21) | -0.09 (1.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.36 (0.99) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Sno (n=67,0,68,0,67,73,73,79,0,66,0) | 3.28 (22.99) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.29 (22.26) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.46 (21.97) | -4.66 (23.46) | -4.11 (21.33) | -4.05 (23.62) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.91 (23.91) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2: Som (n=67,0,68,0,68,73,73,77,0,66,0) | -3.18 (18.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.00 (18.33) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.37 (18.05) | -0.73 (16.20) | -2.74 (15.79) | -3.03 (17.76) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.22 (18.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: SPS (n=62,0,59,0,63,65,63,70,0,61,0) | -5.54 (12.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -10.51 (20.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.97 (18.57) | -2.00 (19.98) | -5.19 (19.19) | -4.62 (17.24) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.95 (18.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: OSP (n=62,0,59,0,63,65,63,69,0,61,0) | -7.27 (11.71) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -11.21 (18.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -5.59 (18.71) | -3.64 (18.32) | -5.63 (17.18) | -6.42 (15.31) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.03 (17.70) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Ade (n=62,0,59,0,63,65,63,70,0,61,0) | 1.45 (22.39) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 11.19 (27.55) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.87 (27.51) | 4.77 (29.32) | 6.51 (25.15) | 6.57 (32.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.82 (23.47) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: ASOB (n=62,0,59,0,63,65,64,70,0,61,0) | -3.87 (24.52) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -7.46 (24.89) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.81 (28.70) | 2.46 (26.10) | -2.81 (23.87) | 1.43 (24.15) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.97 (25.22) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: SD (n=62,0,59,0,63,65,64,70,0,61,0) | -9.74 (16.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -13.43 (22.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -9.25 (23.07) | -6.73 (22.54) | -8.22 (20.59) | -8.45 (18.59) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.97 (21.46) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Opt (n=63,0,59,0,64,65,65,70,0,61,0) | 0.00 (0.54) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.07 (0.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.03 (0.64) | 0.08 (0.62) | -0.05 (0.57) | 0.01 (0.58) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.08 (0.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Qua (n=62,0,57,0,63,65,64,68,0,61,0) | 0.16 (1.43) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 0.40 (1.32) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.73 (8.24) | -0.42 (3.80) | 0.28 (1.52) | 0.74 (5.57) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.33 (9.25) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Sno (n=61,0,59,0,63,65,64,70,0,61,0) | 0.66 (22.20) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -0.34 (27.67) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -2.54 (28.85) | -2.15 (26.25) | 1.56 (24.25) | -1.14 (22.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -3.28 (19.38) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12: Som (n=62,0,59,0,63,65,64,68,0,61,0) | -6.56 (18.60) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -6.33 (19.08) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -1.06 (19.20) | 1.54 (23.06) | -2.81 (20.33) | -4.90 (20.72) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | -4.37 (21.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24: SPS (n=40,20,44,13,55,64,58,52,12,34,17) | -8.25 (15.47) | -0.50 (15.83) | -11.97 (19.23) | -6.92 (18.13) | -4.12 (20.03) | -3.33 (16.38) | -8.62 (18.34) | -7.82 (18.23) | -3.33 (20.84) | -6.27 (19.96) | -2.16 (16.71)
  Week 24: OSP (n=40,20,44,13,55,64,58,51,12,34,17) | -10.18 (14.38) | -2.81 (14.39) | -12.16 (17.87) | -8.50 (16.00) | -6.04 (19.83) | -4.83 (16.17) | -9.82 (16.06) | -9.24 (18.00) | -3.38 (18.83) | -6.01 (18.67) | -1.96 (18.70)
  Week 24: Ade (n=40,20,44,13,55,64,58,52,12,34,17) | 7.75 (26.36) | -6.00 (25.42) | 11.59 (24.30) | 9.23 (23.97) | 8.00 (28.11) | 6.72 (29.33) | 5.52 (26.70) | 11.92 (32.36) | -1.67 (39.73) | -1.18 (29.72) | 8.82 (19.00)
  Week 24: ASOB (n=40,20,44,13,55,64,59,52,12,34,17) | -3.50 (20.20) | -7.00 (29.22) | -11.36 (27.42) | -1.54 (26.41) | -3.27 (24.27) | 0.63 (24.94) | -10.17 (25.56) | -5.38 (19.45) | -6.67 (21.46) | -11.18 (21.57) | 3.53 (26.68)
  Week 24: SD (n=40,20,44,13,55,64,59,52,12,34,17) | -13.66 (18.64) | -6.31 (17.76) | -15.88 (24.63) | -13.75 (21.22) | -6.59 (25.51) | -6.64 (22.53) | -13.98 (18.70) | -8.94 (22.39) | -7.19 (18.41) | -7.06 (23.78) | -1.18 (27.63)
  Week 24: Opt (n=40,20,44,13,55,64,60,53,12,36,17) | 0.00 (0.51) | 0.00 (0.65) | 0.07 (0.62) | -0.08 (0.64) | 0.02 (0.62) | 0.08 (0.65) | -0.05 (0.53) | 0.02 (0.54) | 0.00 (0.74) | -0.08 (0.60) | -0.06 (0.56)
  Week 24: Qua (n=40,20,43,13,55,64,59,51,11,35,17) | -0.10 (1.26) | 0.00 (1.65) | 0.35 (1.56) | 0.38 (1.66) | 0.33 (2.13) | -0.42 (3.97) | 0.31 (1.44) | 0.08 (1.04) | 3.36 (13.89) | 0.29 (1.45) | 0.24 (1.25)
  Week 24: Sno (n=40,19,44,13,54,64,59,52,12,34,17) | 3.50 (25.17) | -1.05 (23.55) | 2.73 (28.48) | 6.15 (18.95) | -7.04 (24.92) | 0.31 (28.84) | 2.37 (22.92) | 1.54 (28.79) | 5.00 (30.90) | -6.47 (26.84) | -1.18 (11.11)
  Week 24: Som (n=40,20,44,13,55,64,59,51,11,34,17) | -5.33 (21.94) | 0.67 (18.34) | -2.58 (20.29) | -4.10 (15.04) | -2.18 (21.08) | -1.04 (20.03) | -6.55 (20.02) | -6.80 (21.19) | -4.24 (18.68) | -7.06 (17.36) | -2.35 (15.45)

30. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale
Description: FACIT-Fatigue scale (FS) is a 13-item questionnaire. Participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-FS score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Week 2, 12, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 70 | 21 | 68 | 13 | 71 | 73 | 75 | 79 | 12 | 69 | 17
units on a scale
  Baseline (n=70,0,68,0,71,73,75,79,0,69,0) | 28.17 (10.50) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 29.92 (11.98) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 28.76 (10.42) | 30.06 (10.85) | 29.48 (10.19) | 29.76 (11.02) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.23 (11.13) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 2 (n=68,0,68,0,68,73,73,78,0,66,0) | 30.41 (12.01) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.65 (10.64) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 32.46 (11.78) | 32.51 (10.58) | 33.41 (10.10) | 33.36 (10.93) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 33.88 (8.90) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=61,0,59,0,63,65,64,69,0,61,0) | 33.25 (10.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.44 (11.16) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 34.30 (10.87) | 33.17 (9.43) | 35.05 (10.17) | 33.99 (11.61) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 35.42 (10.04) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24 (n=39,20,44,13,55,64,59,51,12,35,17) | 36.69 (10.42) | 28.08 (11.07) | 35.48 (11.66) | 34.92 (9.40) | 36.78 (10.75) | 35.36 (10.01) | 36.80 (9.85) | 38.24 (9.46) | 29.50 (12.27) | 37.17 (10.12) | 37.47 (9.87)

31. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale at Week 2, 12 and 24/ET
Description: FACIT-FS is a 13-item questionnaire. Participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-FS score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Week 2, 12, 24/ET
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Number analyzed (Participants) | 68 | 21 | 68 | 13 | 68 | 72 | 73 | 78 | 12 | 66 | 17
units on a scale
  Week 2 (n=68,0,68,0,68,72,73,78,0,66,0) | 1.96 (7.99) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.74 (7.80) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 3.54 (7.71) | 2.80 (7.40) | 3.68 (7.24) | 3.37 (6.56) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 1.61 (6.21) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 12 (n=61,0,59,0,63,65,64,69,0,61,0) | 4.82 (8.53) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 5.79 (10.95) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 4.90 (8.98) | 2.18 (9.25) | 5.41 (9.02) | 4.51 (9.27) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12. | 2.71 (9.94) | NA (NA) — Data not available at this time point since the reassignment to CP-690,550 5 mg was after Week 12.
  Week 24 (n=39,20,44,13,55,64,59,50,12,35,17) | 6.23 (9.66) | 3.73 (10.35) | 5.33 (9.42) | 5.62 (11.57) | 7.18 (9.08) | 4.49 (9.43) | 6.54 (8.90) | 6.88 (9.28) | 4.75 (10.84) | 3.23 (12.13) | 4.18 (6.09)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- CP-690,550 1 mg: CP-690,550 1 mg tablet orally twice daily up to Week 24.
- CP-690,550 1 mg to CP-690,550 5 mg (R): CP-690,550 1 mg tablet orally twice daily up to Week 12 followed by CP-690,550 5 mg tablet orally twice up to Week 24.
- CP-690,550 3 mg: CP-690,550 3 mg tablet orally twice daily up to Week 24.
- CP-690,550 3 mg to CP-690,550 5 mg (R): CP-690,550 3 mg tablet orally twice daily up to Week 12 followed by CP-690,550 5 mg tablet orally twice up to Week 24.
- CP-690,550 5 mg: CP-690,550 5 mg tablet orally twice daily up to Week 24.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily up to Week 24.
- CP-690,550 15 mg: CP-690,550 15 mg tablet orally twice daily up to Week 24.
- CP-690,550 20 mg: CP-690,550 20 mg tablet orally once daily as morning dose and matching placebo tablet orally once daily as evening dose up to Week 24.
- CP-690,550 20 mg to CP-690,550 5 mg (R): CP-690,550 20 mg tablet orally once daily as morning dose and matching placebo tablet orally once daily as evening dose up to Week 12 followed by CP-690,550 5 mg tablet orally twice daily up to Week 24.
- Placebo: Matching placebo tablet orally twice daily up to Week 24.
- Placebo to CP-690,550 5 mg (R): Matching placebo tablet orally twice daily up to Week 12 followed by CP-690,550 5 mg tablet orally twice up to Week 24.
Arm/Group | CP-690,550 1 mg | CP-690,550 1 mg to CP-690,550 5 mg (R) | CP-690,550 3 mg | CP-690,550 3 mg to CP-690,550 5 mg (R) | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | CP-690,550 20 mg | CP-690,550 20 mg to CP-690,550 5 mg (R) | Placebo | Placebo to CP-690,550 5 mg (R)
Serious Adverse Events (participants affected / at risk) | 1/49 | 1/21 | 4/55 | 0/13 | 4/71 | 1/74 | 6/75 | 4/67 | 0/13 | 0/51 | 0/18
Other Adverse Events (participants affected / at risk) | 28/49 | 14/21 | 30/55 | 10/13 | 40/71 | 45/74 | 46/75 | 37/67 | 6/13 | 29/51 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 1 mg (N=49) | CP-690,550 1 mg to CP-690,550 5 mg (R) (N=21) | CP-690,550 3 mg (N=55) | CP-690,550 3 mg to CP-690,550 5 mg (R) (N=13) | CP-690,550 5 mg (N=71) | CP-690,550 10 mg (N=74) | CP-690,550 15 mg (N=75) | CP-690,550 20 mg (N=67) | CP-690,550 20 mg to CP-690,550 5 mg (R) (N=13) | Placebo (N=51) | Placebo to CP-690,550 5 mg (R) (N=18)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dissociative disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 1 mg (N=49) | CP-690,550 1 mg to CP-690,550 5 mg (R) (N=21) | CP-690,550 3 mg (N=55) | CP-690,550 3 mg to CP-690,550 5 mg (R) (N=13) | CP-690,550 5 mg (N=71) | CP-690,550 10 mg (N=74) | CP-690,550 15 mg (N=75) | CP-690,550 20 mg (N=67) | CP-690,550 20 mg to CP-690,550 5 mg (R) (N=13) | Placebo (N=51) | Placebo to CP-690,550 5 mg (R) (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual disturbance (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 1 | 2 | 1 | 0 | 1 | 3 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 1 | 1 | 1 | 9 | 1 | 3 | 1 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 1 | 3 | 5 | 4 | 2 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 3 | 1 | 2 | 4 | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 1 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 4 | 2 | 1 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 1 | 2 | 5 | 3 | 1 | 1 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 1 | 5 | 2 | 6 | 4 | 1 | 3 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 3 | 1 | 2 | 0 | 1 | 2 | 1 | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 3 | 5 | 5 | 2 | 4 | 2 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 2 | 5 | 4 | 5 | 6 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 5 | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 2 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Electrocardiogram ST-T change (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cluster headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 2 | 2 | 3 | 4 | 9 | 3 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 3 | 6 | 2 | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpable purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 2 | 4 | 2 | 1 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 2 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 1
Venous stasis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.